# ANALYSIS DISPLAY PLAN

TABLE and LISTING MOCK-UPs

Compound: PHA-848125AC Protocol No.: CDKO-125a-007

Protocol title: Phase II Study of Oral PHA-848125AC in Patients with Malignant Thymoma Previously Treated with Multiple Lines of

Chemotherapy

Clinical phase: Phase II

Author: Vincenzo Pace, Biostatistics

| GENERAL ISSUES | 8 |
|---|---|
| APPENDIX 1: STUDY INFORMATION | 9 |
| Appendix 1 – Section 9 – Statistical and Analytical Issues | 10 |
| Appendix 1.9.1. <x> – Treatment Efficacy - Kaplan Meier Estimates for Progression Free Survival – Treated / Evaluable Patients –</x> | |
| Appendix 1.9.2. <x> - Treatment Efficacy - Kaplan Meier Estimates for Overall Survival - Treated / Evaluable Patients</x> | 11 |
| $Appendix \ 1.9.3. < x > - \ Treatment \ Efficacy \ - \ Kaplan \ Meier \ Estimates \ for \ Duration \ of \ Response \ - \ Treated \ / \ Evaluable \ Patients \ - \dots -$ | 12 |
| APPENDIX 2: SUMMARY TABLES | 13 |
| Appendix 2 - Section 1 - Patient Disposition | 14 |
| Appendix 2.1.1 - Patient Disposition: Patient Screening - Screened Patients – | |
| Appendix 2.1.2 - Patient Disposition: Patient Disposition by Investigational Site - Enrolled Patients – | 15 |
| Appendix 2.1.3 - Patient Disposition: Study Period Completion and Primary Off Study Reason - Enrolled Patients - | |
| Appendix 2.1.4 - Patient Disposition: Treatment Period Completion and Primary Off Treatment Reason - Treated Patients | |
| Appendix 2.1.5 – Patient Disposition: Frequency of Patients according to Time on Treatment - Treated Patients – | 18 |
| Appendix 2 – Section 2 – Demography and Pretreatment Characteristics | 19 |
| Appendix 2.2.1 – Demography and Pretreatment: Demography Characteristics - Treated Patients - | |
| Appendix 2.2.2 – Demography and Pretreatment: Summary Statistics of Age, Weight and Height - Treated Patients - | |
| Appendix 2.2.3 – Demography and Pretreatment: Tumor History - Primary Diagnosis and Diagnosis at Study Entry - Treated Patients – | |
| Appendix 2.2.4 – Demography and Pretreatment: Tumor History – Time from Primary Diagnosis and Diagnosis at Study Entry to Treatment | |
| Start - Treated Patients - | |
| Appendix 2.2.5 – Demography and Pretreatment: History of Other Cancers - Treated Patients | |
| Appendix 2.2.6 - Demography and Pretreatment: Tumor History - Prior Antitumor Treatments / Procedures: Type and Setting - Treated I | |
| Appendix 2.2.7 – Treatment Efficacy: Oncologic Assessment at Study Entry - Treated Patients – | |
| Appendix 2.2.8 – Demography and Pretreatment: Signs and Symptoms - Treated Patients - | |
| Appendix 2 – Section 3 – Treatment Exposure | |
| Appendix 2.3.1 – Treatment Exposure: Summary Statistics of the Number of Cycles / Weeks of Treatment - Treated Patients | |
| Appendix 2.3.2 - Treatment Exposure: Frequency Distribution of Cycles according to the Percentage of Scheduled Dose Administered - T | |
| Patients | 28 |

| Appendix 2.3.3 – Treatment Exposure: Summary Statistics of Dose Intensity, Relative Dose Intensity and Cumulative Dose - Whole Treatment | nt |
|---|---|
| Period Treated Patients - | |
| Appendix 2.3.4 - Treatment Exposure: Frequency Distribution of Cycles according to their Duration - Treated Patients – | 30 |
| Appendix 2.3.5 – Treatment Exposure: Frequency Distributions of Patients and Cycles with Treatment Modifications - Treated Patients | 31 |
| Appendix 2.3.6 – Treatment Exposure: Frequency Distributions of Patients by Reasons for Treatment Modifications - Treated Patients – | |
| Appendix 2 – Section 4 – Treatment Efficacy | 33 |
| Appendix 2.4.1. <x> – Treatment Efficacy: Progression Free Survival Rate at 3 Months - Evaluable Patients/Treated –</x> | 33 |
| Figure 2.4.1. <x> – Treatment Efficacy: Kaplan-Meier Curve for Progression Free Survival - Evaluable Patients/Treated –</x> | 34 |
| Appendix 2.4.2. <x> – Treatment Efficacy: Best Confirmed Tumor Response - Evaluable/Treated</x> | 35 |
| Appendix 2.4.3. <x> – Treatment Efficacy: Best Unconfirmed Tumor Response - Evaluable/Treated -</x> | |
| Appendix 2.4.4. <x> – Treatment Efficacy: Statistical Analysis of Time-To-Event Endpoints - Treated / Evaluable Patients</x> | |
| Appendix 2.4.4. <x> – Treatment Efficacy: Statistical Analysis of Time-To-Event Endpoints - Treated / Evaluable Patients</x> | 37 |
| Figure 1.9.2. <x> – Treatment Efficacy: Kaplan-Meier Curve for Overall Survival - Treated / Evaluable Patients–</x> | 38 |
| Appendix 2.4.5 – Treatment Efficacy: ECOG Performance Status: On Treatment Worst Assessment vs. Pretreatment - Treated Patients with a | |
| Least One Assessment On Treatment - | 39 |
| Appendix 2 – Section 5 – Adverse Events | 40 |
| Appendix 2.5.1 – Adverse Events: Patients with on Treatment AEs by System Organ Class and Maximum CTC Grade - Treated Patients – Appendix 2.5.2 – Adverse Events: Patients with on Treatment AEs by AE MedDRA Preferred Term and Maximum CTC Grade - Treated | 40 |
| Patients – Patients – CTG G. 1. T | |
| Appendix 2.5.3 – Adverse Events: Patients with on Treatment AEs by SOC, AE MedDRA Preferred Term and Maximum CTC Grade - Treate Patients - | |
| Appendix 2.5.4 – Adverse Events: Patients with AEs with Possible to Definite Relationship to Study Treatment by SOC and Maximum CTC | |
| | 43 |
| Appendix 2.5.5 – Adverse Events: Patients with AEs with Possible to Definite Relationship to Study Treatment by AE MedDRA Preferred Te and Maximum CTC Grade - Treated Patients – | |
| Appendix 2.5.6 - Adverse Events: Patients with AEs with Possible to Definite Relationship to Study Treatment by SOC, AE MedDRA Prefer | red |
| Term and Maximum CTC Grade - Treated Patients – | 45 |
| Appendix 2.5.7 - Adverse Events: Patients with on Treatment Serious AEs by SOC, AE MedDRA Preferred Term and Maximum CTC Grade | e - |
| Treated Patients – | |
| Appendix 2.5.8 – Adverse Events: Patients with Serious AEs with Possible to Definite Relationship to Study Treatment by SOC, AE MedDR. | |
| Preferred Term and Maximum CTC Grade - Treated Patients – | 47 |

| Appendix 2.5.9 – Adverse Events: Patients with on Treatment AEs Leading to Withdrawal from Study Treatment by SOC, AE MedDRA | 40 |
|---|---|
| Preferred Term and Maximum CTC Grade - Treated Patients – | |
| Appendix 2 - Section 6 – Laboratory Assessments | |
| Appendix 2.6.1 – Hematology: Frequency Distribution of Patients based on Maximum CTC Grade On Treatment versus Pretreatment - Treat | ed |
| Patients with at Least One Assessment On Treatment All Cycles, Cycle 1, Cycles > 1- | |
| Appendix 2.6.2 – Hematology: Frequency Distribution of Treatment Cycles based on Maximum CTC Grade On Treatment versus Pretreatment | |
| Cycles with at Least One Assessment All Cycles, Cycle 1, Cycles > 1 - | |
| Appendix 2.6.3 - Blood Chemistry: Frequency Distribution of Patients based on Maximum CTC Grade On Treatment versus Pretreatment (P | |
| I) - Treated Patients with at Least One Assessment On Treatment All Cycles, Cycle 1, Cycles > 1- | |
| Appendix 2.6.4 – Blood Chemistry: Frequency Distribution of Patients based on Maximum CTC Grade On Treatment versus Pretreatment (P | |
| II) - Treated Patients with at Least One Assessment On Treatment All Cycles - | 53 |
| Appendix 2.6.5 – Blood Chemistry: Frequency Distribution of Treatment Cycles based on Maximum CTC Grade On Treatment versus | <i>E 1</i> |
| Pretreatment (Part I) - Cycles with at Least One Assessment All Cycles, Cycle 1, Cycles > 1 | 54 |
| Pretreatment (Part II) - Cycles with at Least One Assessment All Cycles- | 55 |
| Appendix 2.6.7 – Coagulation: Frequency Distribution of Patients based on Maximum CTC Grade On Treatment versus Pretreatment - Treatment - | 55<br>ed |
| Patients with at Least One Assessment On Treatment All Cycles, Cycle 1, Cycles > 1 - | |
| Appendix 2.6.8 – Laboratory Tests without a NCI-CTC Grade: Frequency Distribution of Patients Based on On Treatment Worst Assessment | |
| versus Pretreatment - Treated Patients with at Least One Assessment On Treatment All Cycles, Cycle 1, Cycles > 1 | 57 |
| Appendix 2.7 – Other Safety Assessments | 58 |
| Appendix 2.7.1 – Other Safety Assessments: Blood Pressure - On Treatment Worst Assessment versus Pretreatment - Treated Patients with a | t |
| Least One Assessment On Treatment - | |
| Appendix 2.7.2 – Other Safety Assessments: ECG - On Treatment Assessment versus Pretreatment Condition - Treated Patients with at Least | |
| One Assessments On Treatment - | |
| Appendix 2.7.3 – Other Safety Assessments: ECG - On Treatment Abnormality Findings - Treated Patients with at Least One Assessment Or Treatment – | |
| Appendix 2.7.4 – Other Safety Assessments: Funduscopic Examination - On Treatment Worst Assessment versus Pretreatment - Treated Pati | |
| with at Least One Assessment On Treatment - | |
| APPENDIX 3: INDIVIDUAL DATA LISTINGS | 62 |
| Appendix 3 - Section 1 - Patient Disposition | 63 |
| rr | |

| Appendix 3.1.1 – Patient Disposition: Patient Registration – Registered Patients – | 63 |
|---|---|
| Appendix 3.1.2 – Patient Disposition: Registered but Not Enrolled Patients - Screening Failures - | |
| Appendix 3.1.3 – Patient Disposition: Summary of Patient Information - Enrolled Patients- | |
| Appendix 3.1.4 – Patient's Survival Status during Follow Up - Treated Patients- | |
| Appendix 3 - Section 2 - Protocol Deviations | 67 |
| Appendix 3.2.1 - Protocol Deviations: Violations of Inclusion / Exclusion Criteria - Enrolled Patients – | 67 |
| Appendix 3 – Section 3 – Patients Evaluability for Efficacy Analysis | 68 |
| Appendix 3.3.1 –Evaluability for Efficacy Analysis: Evaluability Criteria and Individual Evaluability Status - Enrolled Patients- | |
| Appendix 3 – Section 4 – Demography and Pretreatment | |
| Appendix 3.4.1 - Demography and Pretreatment: Tumor History - Primary Diagnosis - Treated Patients | 69 |
| Appendix 3.4.2 - Demography and Pretreatment: Tumor History – Diagnosis at Study Entry - Treated Patients – | 70 |
| Appendix 3.4.3 - Demography and Pretreatment: Tumor History – NCI Confirmation of Diagnosis - Treated Patients – | 71 |
| Appendix 3.4.4 - Demography and Pretreatment: History of Other Cancers - Treated Patients- | 72 |
| Appendix 3.4.5 - Demography and Pretreatment: Tumor History - Prior Antitumor Treatments/Procedures - Treated Patients | 73 |
| Appendix 3.4.6 - Demography and Pretreatment: Tumor History - Prior Systemic Therapies - Treated Patients – | |
| Appendix 3.4.7 – Demography and Pretreatment: Tumor History - Prior Surgeries - Treated Patients – | 75 |
| Appendix 3.4.8 – Demography and Pretreatment: Tumor History - Prior Radiotherapies - Treated Patients – | 76 |
| Appendix 3.4.9 - Demography and Pretreatment: General Medical History and Physical Examination Findings - Treated Patients | 77 |
| Appendix 3 – Section 5 – Treatment Exposure | 78 |
| Appendix 3.5.1 – Treatment Exposure: Treatment Administration Details - Treated Patients – | 78 |
| Appendix 3.5.2 – Treatment Exposure: Reasons for Treatment Delay, Dose Reduction - Treated Patients | 79 |
| Appendix 3.5.3 – Treatment Exposure: Dose Intensity and Cumulative Dose - Treated Patients – | 80 |
| Appendix 3.5.4 – Treatment Exposure: Pharmacokinetics Blood Sampling Time - Treated Patients – | 81 |
| Appendix 3 – Section 6 – Treatment Efficacy | 82 |
| Appendix 3.6.1 - Treatment Efficacy - Target and Non Target Lesions by Assessment Visit - Treated Patients | 82 |
| Appendix 3.6.2 - Treatment Efficacy - Response Status by Assessment Visit - Treated Patients - | 83 |
| Appendix 3.6.3 - Treatment Efficacy – Best Overall Response and Time to Progression, Progression Free Survival, Overall Survival, Respon Duration and Stable Disease Duration - Treated Patients - | |
| Appendix 3.6.4 – Treatment Efficacy: ECOG Performance Status - Treated Patients - | |
| Appendix 3 – Section 7 – Adverse Events | |
| 11ppendia v Svedon / 11croise Divinguismussimusmussimusmusmusmusmusmusmusmusmusmusmusmusmusm | 00 |

| Appendix 3.7.1 – Adverse Events: All Reported Adverse Events by Assessment Visit and AE MedDRA Preferred Term - Treated Patients | s 86 |
|---|---|
| Appendix 3.7.2 - Adverse Events: Adverse Events Related to Study Procedure at Pretreatment - Treated Patients – | 87 |
| Appendix 3.7.3 – Adverse Events: Serious Adverse Events - Treated Patients - | 88 |
| Appendix 3.7.4 – Adverse Events: Adverse Events with CTC Grade 3 to 5 - Treated Patients - | |
| Appendix 3.7.5 – Adverse Events: Patients with Adverse Events Leading to Withdrawal from Study Treatment - Treated Patients | |
| Appendix 3.7.6 – Adverse Events: End of AE Reporting Period and Follow-Up - Treated Patients – | |
| Appendix 3.7.7 – Adverse Events: All Reported Adverse Events by System Organ Class, AE MedDRA Preferred Term and Investigator's | |
| Treated Patients - | |
| Appendix 3.7.8 – Adverse Events: Hospitalization - Treated Patients - | 93 |
| Appendix 3.7.9 – Deaths - Treated Patients - | |
| Appendix 3.7.10 – Deaths: Autopsy Result - Treated Patients – | 95 |
| Appendix 3 - Section 8 – Laboratory Assessments | 96 |
| Appendix 3.8.1 – Laboratory Assessments: Hematology by Laboratory Test, Patient and Study Period - Treated Patients | |
| Appendix 3.8.2 – Laboratory Assessments: Blood Chemistry by Laboratory Test, Patient and Study Period - Treated Patients | |
| Appendix 3.8.3 – Laboratory Assessments: Coagulation by Patient, Study Period and Laboratory Test - Treated Patients – | 98 |
| Appendix 3.8.4 – Laboratory Assessments: Urinalysis - Treated Patients – | |
| Appendix 3.8.5 – Laboratory Assessments: Laboratory Normal Ranges of Hematological Tests | |
| Appendix 3.8.6 – Laboratory Assessments: Laboratory Normal Ranges of Non-Hematological Tests - Treated Patients - | 101 |
| Appendix 3 - Section 9 - Other Safety Assessments | 102 |
| Appendix 3.9.1 – Other Safety Assessments: Vital Signs - Treated Patients – | |
| Appendix 3.9.2 – Other Safety Assessments: ECG - Treated Patients – | |
| Appendix 3.9.3 – Other Safety Assessments: Visual Acuity and Funduscopic Examination - Treated Patients – | 104 |
| Appendix 3.9.4 – Other Safety Assessments: Chest X-Ray - Treated Patients – | 105 |
| Appendix 3.9.5 – Other Safety Assessments: Pregnancy Test - Treated Patients – | 106 |
| Appendix 3.9.6 – Other Safety Assessments: Physical Examination - Treated Patients - | 107 |
| Appendix 3 – Section 10 – Other Information | 108 |
| Appendix 3.10.1 - Other Information: Concomitant Medications - Treated Patients – | 108 |
| Appendix 3.10.2 – Other Information: Concomitant Radiotherapies - Treated Patients – | 109 |
| Appendix 3.10.3 – Other Information: Blood Derivatives - Treated Patients - | |
| Appendix 3.10.4 - Other Information: Other Anti-Tumor Therapies at Follow-up - Treated Patients – | |
| Appendix 3.10.5 - Other Information: Physician's Comments - Treated Patients - | 112 |

| ADDITIONAL DISPLAYS | . 113 |
|---|---|
| Listing 3.3.1 – Patients Evaluability for Efficacy Analysis: Patients not Included in the Efficacy Analysis of Evaluable Patients - Enrolled | |
| Patients | |
| Listing 3.4.1 – Demography and Pretreatment: Tumor History - Summary of Prior Antitumor Treatment Procedure - Treated Patients – | . 115 |
| Listing 3.7.1 - Adverse Events: All Reported Adverse Events by AE MedDRA Preferred Term and Assessment Visit - Treated Patients – | . 116 |
| Listing 3.7.2 – Adverse Events: AEs with Possible/Probable/Definite Relationship to Study Treatment - Treated Patients | . 117 |
| Listing 3.7.3 – Adverse Events: AEs Leading to Dose Delay or Change - Treated Patients - | . 118 |
| Listing 3.8.1 - Laboratory Assessments: Hematology by Patient, Study Period and Laboratory Test - Treated Patients - | . 119 |
| Lisring 3.8.2 - Laboratory Assessments: Hematology by Laboratory Test, Patient and Study Periods with More than One Assessment - Treate | ed |
| Patients - | |
| Listing 3.8.3 – Laboratory Assessments: Hematology – Maximum CTC Grade by Laboratory Test, Patient and Time Window - Treated Patient | nts – |
| | . 121 |
| Listing 3.8.4 - Laboratory Assessments: Blood Chemistry by Patient, Study Period and Laboratory Test - Treated Patients – | . 122 |
| Listing 3.8.5 – Laboratory Assessments: Blood Chemistry by Laboratory Test, Patient and Study Periods with More than One Assessment - | |
| Treated Patients - | . 123 |
| Listing 3.8.6 – Laboratory Assessments: Blood Chemistry - Maximum CTC Grade by Laboratory Test, Patient and Time Window (Part I) - | |
| Treated Patients - | . 124 |
| Listing 3.8.7 – Laboratory Assessments: Blood Chemistry - Maximum CTC Grade by Laboratory Test, Patient and Time Window (Part II) - | |
| Treated Patients - | . 125 |
| REVISION HISTORY | . 126 |
| : : _ : _ : _ : _ : _ : _ : _ : | 0 |

#### **GENERAL ISSUES**

"Page by Regimen" for outputs, in this study one regimen only: 150 mg/day x 7 days q 2 wks.

The outputs will have names starting with "Appendix 1.9.n.<X>" or "Appendix 2.4.n.<X>" or "Figure 2.4.n.<X>", where X will be set to different values according to the subset population described: <x> = 1 for evaluable patients, 2 for treated patients.

**APPENDIX 1: STUDY INFORMATION** 

# Appendix 1 – Section 9 – Statistical and Analytical Issues

Appendix 1.9.1.<x> – Treatment Efficacy - Kaplan Meier Estimates for Progression Free Survival – Treated / Evaluable Patients –

#### Page by Regimen

| Progression Free<br>Survival<br>(days) | Pat No | Number of Patients Failed | Number of Patients<br>Left | Probability | Standard Error | 95% CI – LL (**) | 95% CI – UL (**) |
|---|---|---|---|---|---|---|---|
| 0 | 008 | XX | XX | 1 | 0.xxx | 0.xx | 0.xx |
| 1 * | | XX | XX | 0.xx | 0.xxx | 0.xx | 0.xx |

[Protocol No.; Study Description]

[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Descriptive statistics are obtained with SAS PROC LIFETEST considering the Kaplan-Meier method. For Pat-No use ID statement in PROC LIFETEST

<sup>\*</sup> Censored Observation

<sup>\*\*</sup> Confidence Intervals around Kaplan Meier estimates

# Appendix 1.9.2. < x > - Treatment Efficacy - Kaplan Meier Estimates for Overall Survival - Treated / Evaluable Patients -

# Page by Regimen

| Overall Survival (months) | Pat No | Number of Patients<br>Failed | Number of Patients<br>Left | Probability | Standard Error | 95% CI – LL (**) | 95% CI – UL (**) |
|---|---|---|---|---|---|---|---|
| 0 | 011 | XX | XX | 1 | 0.xxx | 0.xx | 0.xx |
| 1 * | •••• | XX | XX | 0.xx | 0.xxx | 0.xx | 0.xx |


[Program Path; Date/Time Produced; Date Data Extract]

# **Programming Notes:**

Descriptive statistics are obtained with SAS PROC LIFETEST considering the Kaplan-Meier method. For Pat-No use ID statement in PROC LIFETEST

<sup>\*</sup> Censored Observation

<sup>\*\*</sup> Confidence Intervals around Kaplan Meier estimates

# Appendix 1.9.3.<x > - Treatment Efficacy - Kaplan Meier Estimates for Duration of Response - Treated / Evaluable Patients -

# Page by Regimen

| Duration of<br>Response<br>(days) | Pat-No | Number of Patients<br>Failed | Number of Patients<br>Left | Probability | Standard Error | 95% CI – LL (**) | 95% CI – UL (**) |
|---|---|---|---|---|---|---|---|
| 0 | | XX | XX | 1 | 0.xxx | 0.xx | 0.xx |
| 1 * | | XX | XX | 0.xx | 0.xxx | 0.xx | 0.xx |


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Descriptive statistics are obtained with SAS PROC LIFETEST considering the Kaplan-Meier method. For Pat-No use ID statement in PROC LIFETEST

<sup>\*</sup> Censored Observation

<sup>\*\*</sup> Confidence Intervals around Kaplan Meier estimates

**APPENDIX 2: SUMMARY TABLES** 

# Appendix 2 - Section 1 - Patient Disposition

Appendix 2.1.1 - Patient Disposition: Patient Screening - Screened Patients -

| | n | % |
|------------------------------------|-----|-------|
| Total Patients Screened | XXX | 100.0 |
| Patients Screened and not Enrolled | XXX | XXX.X |
| Patients Enrolled | XXX | XXX.X |

%=(n/Total patients screened)\*100


Appendix 2.1.2 - Patient Disposition: Patient Disposition by Investigational Site - Enrolled Patients -

| | | Enrolled Patients | | |
|---|---|---|---|---|
| | | All Enrolled Treated Not Treat | | |
| | | (N=xx) | (N=xx) | (N=xx) |
| | n | | | n |
| Investigational Site | All Centers | XX | XX | XX |
| | <center_1></center_1> | XX | XX | XX |
| | <center_2></center_2> | XX | XX | XX |

Treated / Not Treated: patients who received / did not receive at least one treatment dose


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

N=xx: xx is the total number of patients for each distinct patient group (treated, not treated, all enrolled)

Appendix 2.1.3 - Patient Disposition: Study Period Completion and Primary Off Study Reason - Enrolled Patients -

| | | | Enrolled Patients | | | | |
|---|---|---|---|---|---|---|---|
| | | All Er | All Enrolled Treated (N=xx) (N=xx) | | ated | Not T | reated |
| | | (N= | | | xx) | (N=xx) | |
| | | n | % | n | % | n | % |
| Off Study Patients | Total Off Study | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Death | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Lost to follow-up | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | ••• | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Reason Not Provided | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| On Study Patients | Total On Study | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Off Treatment | XX | XXX.X | XX | XXX.X | | |

%=(n/N)\*100

On Study Patients: patients whose Off Study Reason form has not been received and no death is reported.


[Program Path; Date/Time Produced; Date Data Extract]

# **Programming Notes:**

N=xx: xx is the total number of patients for each analyzed group (treated, not treated, all enrolled)

Appendix 2.1.4 - Patient Disposition: Treatment Period Completion and Primary Off Treatment Reason - Treated Patients -

| | | | l Patients<br>=xx) |
|---|---|---|---|
| | | n | % |
| Off Treatment Patients | Total Off Treatment | XXX | XXX.X |
| | Adverse Event Lack of Compliance | XXX | XXX.X |
| | | XXX | XXX.X |
| | | XXX | XXX.X |
| | Reason Not Provided | XXX | XXX.X |
| On Treatment Patients | Still on Treatment | XXX | XXX.X |

%=(n/N)\*100

On Treatment Patients: patients whose last available information refers to the study treatment period.


Appendix 2.1.5 – Patient Disposition: Frequency of Patients according to Time on Treatment - Treated Patients –

| Time on Treatment | Treated Patients (N=xx) | |
|---------------------------|-------------------------|------|
| | n | % |
| Lessor equal to 2 weeks | XX | XX.X |
| > 2 - <u>&lt;</u> 6 weeks | XX | XX.X |
| $> 6 - \le 12$ weeks | XX | XX.X |
| > 12 - ≤18 weeks | XX | XX.X |
| >_18 weeksr | XX | XX.X |

%=(n/N)\*100

Time on Treatment: from first dose date to last dose date.


# Appendix 2 – Section 2 – Demography and Pretreatment Characteristics

Appendix 2.2.1 – Demography and Pretreatment: Demography Characteristics - Treated Patients -

Page by Regimen

| | | | Patients =xx) |
|-------------|----------------|----|---------------|
| | | n | % |
| Gender | Male | XX | XX.X |
| | Female | XX | XX.X |
| | Total Reported | XX | XX.X |
| Race | White | XX | XX.X |
| | | XX | XX.X |
| | Total Reported | XX | XX.X |
| Age (years) | <40 yrs | XX | XX.X |
| | 40 - 54 yrs | XX | XX.X |
| | 55 – 65 yrs | XX | XX.X |
| | > 65 yrs | XX | XX.X |
| | Total Reported | XX | XX.X |

%=(n/N)\*100


Appendix 2.2.2 – Demography and Pretreatment: Summary Statistics of Age, Weight and Height - Treated Patients -

Page by Regimen

| | | Treated Patients |
|-------------|------------|------------------|
| | 1 | (N=xx) |
| Age (years) | No. of Pts | XX |
| | Mean | XX.X |
| | SD | XX.X |
| | Median | XX |
| | Min | XX |
| | Max | XX |
| Weight (Kg) | No. of Pts | XX |
| | Mean | XX.X |
| | SD | XX.X |
| | Median | XX |
| | Min | XX |
| | Max | XX |
| Height (cm) | No. of Pts | XX |
| | Mean | XX.X |
| | SD | XX.X |
| | Median | XX |
| | Min | XX |
| | Max | XX |


Appendix 2.2.3 – Demography and Pretreatment: Tumor History - Primary Diagnosis and Diagnosis at Study Entry - Treated Patients –

#### Page by Regimen

| | | Treated Patients (N=xx) | |
|---|---|---|---|
| | | n | % |
| Primary Diagnosis made by: | Histological | XX | XXX.X |
| | Cytological | XX | XXX.X |
| | Total Reported | XX | XXX.X |
| WHO Classification | B3 – Well Differenciated Thymic Carcinoma | XX | XXX.X |
| | C – Thymic Carcinoma | XX | XXX.X |
| | Total Reported | XX | XXX.X |
| Tumor Extent at Study Entry | Locally Advanced | XX | XXX.X |
| | Metastatic | XX | XXX.X |
| | Total Reported | XX | XXX.X |
| Metastatic Disease Sites | Liver | XX | XXX.X |
| | Other | XX | XXX.X |
| | Total Reported | XX | XXX.X |
| Total No. of Recurrence(s)/Progression(s) | 1 | XX | XXX.X |
| | 2 | XX | XXX.X |
| | >2 | XX | XXX.X |
| | Total Reported | XX | XXX.X |
| Masaoka Clinical Staging at Study Entry | I | XX | XX |
| | IIA | XX | XX |
| | IIB | XX | XX |
| | IIIA | XX | XX |
| | IIIB | XX | XX |
| | IVA | XX | XX |
| | IVB | XX | XX |
| | Total Reported | XX | XXX.X |

#### %=(n/N)\*100

Metastatic Disease Site: pts with more than 1 metastatic site are counted for each reported site. Total reported: no. of pts. independently of the sites involved [Protocol No.; Study Description]

Appendix 2.2.4 – Demography and Pretreatment: Tumor History – Time from Primary Diagnosis and Diagnosis at Study Entry to Treatment Start - Treated Patients –

#### Page by Regimen

| | Treated Patients (N=xx) | | | |
|---|---|---|---|---|
| | No. of<br>Pts. | Min | Median | Max |
| Primary Diagnosis (Months) | XX | XXX.X | XXX.X | XXX.X |
| Current Diagnosis of locally advanced or metastatic disease (Weeks) | XX | XXX.X | XXX.X | XXX.X |


Appendix 2.2.5 – Demography and Pretreatment: History of Other Cancers - Treated Patients -

Page by Regimen

| Previous History of Other Cancers | Treated Patients (N=xx) | |
|-----------------------------------|-------------------------|-------|
| | n | % |
| Yes | XX | XXX.X |
| No | XX | XXX.X |
| Total Reported | XX | XXX.X |

%=(n/N)\*100

[Protocol No.; Study Description] [Program Path; Date/Time Produced; Date Data Extract]

Appendix 2.2.6 - Demography and Pretreatment: Tumor History - Prior Antitumor Treatments / Procedures: Type and Setting - Treated Patients -

# Page by Regimen

| | | | Patients =xx) |
|---|---|---|---|
| | | n % | |
| Prior Antitumor Treatments / Procedures | No prior treatments / procedures | XX | XXX.X |
| | At least one prior treatment / procedure | XX | XXX.X |
| | Total Reported | XX | XXX.X |
| Туре | Surgery only | XX | XXX.X |
| | Systemic only | XX | XXX.X |
| | Radiotherapy only | XX | XXX.X |
| | Surgery + Systemic | XX | XXX.X |
| | | XX | XXX.X |
| Setting | Neo-Adjuvant | XX | XXX.X |
| | Adjuvant | XX | XXX.X |
| | Primary Tumor | XX | XXX.X |
| | | XX | XXX.X |

%=(n/N)\*100


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Type: Count each pt for each tr. / procedure type (e.g. surgery,...) reported, regardless of how many times the same type of tr. is reported for him. Ex.: A pt with systemic reported 3 times and surgery reported 2 times, will be counted once for "systemic + surgery" in the table.

Setting: Count each pt for each reported setting (e.g. neo-adjuvant,...) regardless of how many times the same setting is reported for him. Ex.: A pt with primary tumor reported once and metastatic reported 3 times, will be counted once for primary tumor and once for metastatic.

# Appendix 2.2.7 – Treatment Efficacy: Oncologic Assessment at Study Entry - Treated Patients –

# Page by Regimen

| Tumor Lesions | Treated Pati<br>(N= xx) | |
|---|---|---|
| | n | % |
| Total Reported | XX | XXX.X |
| Patients with Both Target and Non-Target Lesions | XX | XXX.X |
| Target Lesions only | XX | XXX.X |
| Non-Target Lesions only | XX | XXX.X |

%=(n/N)\*100

Tumor Lesions include Lymph Nodes


Appendix 2.2.8 – Demography and Pretreatment: Signs and Symptoms

- Treated Patients -

Page by Regimen

| Treated Patients (N=xx) | | Maximum CTC Grade | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Any | Grade | 3 | -4 | | 1 | | ••• | U | <sup>J</sup> nk |
| System Organ Class | Preferred Term | n % n % | | n | % | n | % | n | % | | |
| Any System | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC 1] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event i | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | ••• | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC i] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Within each by group, SOC and AE (i.e. for each Preferred Term), count patients according to the maximum CTC grade reported for that event and sort SOCs by descending frequency of "Any Term" at "Any Grade".

# Appendix 2 – Section 3 – Treatment Exposure

Appendix 2.3.1 – Treatment Exposure: Summary Statistics of the Number of Cycles / Weeks of Treatment - Treated Patients -

Page by Regimen

| | | Sum.of | | | |
|--------------------|----------|--------------|------|--------|------|
| | No. of | Cycles/Weeks | | | |
| Treatment Duration | Patients | of Treatment | Min | Median | Max |
| Cycles | XX | XX.X | XX.X | XX | XX.X |
| Weeks | XX | XX.X | XX.X | XX | XX.X |

Treatment Duration: from the first dose date to end of treatment.


Appendix 2.3.2 - Treatment Exposure: Frequency Distribution of Cycles according to the Percentage of Scheduled Dose Administered - Treated Patients -

# Page by Regimen

| | | Dose Administered (as Percentage of the Scheduled Dose) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Full | Dose | 80% - < ] | Full Dose | 50% - < 80% | | <50% | |
| No. of | Total No. | No. of | | No. of | | No. of | | No. of | |
| Patients | of Cycles | Cycles | % | Cycles % | | Cycles | % | Cycles | % |
| XX | XXX | XX | XX.X | | | | | | |

Scheduled Dose: assigned dose level (mg/day)\*7, where 7 is the per protocol no. of drug administrations per cycle.

Full Dose: greater or equal 95% of Scheduled Dose


Appendix 2.3.3 – Treatment Exposure: Summary Statistics of Dose Intensity, Relative Dose Intensity and Cumulative Dose

- Whole Treatment Period 
- Treated Patients -

# Page by Regimen

| | Dose Intensity | | | Relative Dose Intensity | | | Cumulative Dose | | |
|---|---|---|---|---|---|---|---|---|---|
| No. | (mg/wk) | | | (%) | | | (mg) | | |
| of Pts | Min | Median | Max | Min | Median | Max | Min | Median | Max |
| XX | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |

Relative Dose Intensity: the ratio between dose intensity and intended dose intensity x 100.


[Program Path; Date/Time Produced; Date Data Extract]

# **Programming Notes:**

The whole stydy period is to be considered for the analysis.

Appendix 2.3.4 - Treatment Exposure: Frequency Distribution of Cycles according to their Duration - Treated Patients -

Page by Regimen

| | | Cycle Duration | | | |
|---|---|---|---|---|---|
| No. of | Total No. | < 13 Days | 13-15 Days | 16-28 Days | > 28 Days |
| Patients | of Cycles | No. of Cycles | No. of Cycles | No. of Cycles | No. of Cycles |
| XX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XXX | XXX | XXX | XXX |


Appendix 2.3.5 – Treatment Exposure: Frequency Distributions of Patients and Cycles with Treatment Modifications - Treated Patients -

#### Page by Regimen

| Treated Patients (N=xx) | No. of I | Patients | No. of Cycles |
|--------------------------|----------|----------|---------------|
| Treatment Modifications | n | % | n |
| Any Modification | XX | XXX.X | XX |
| | XX | XXX.X | XX |
| | XX | XXX.X | XX |
| Intra Cycle Modification | XX | XXX.X | XX |
| | XX | XXX.X | XX |
| | XX | XXX.X | XX |
| Treatment Delay | XX | XXX.X | XX |
| | XX | XXX.X | XX |
| | XX | XXX.X | XX |
| Dose Reduction | XX | XXX.X | XX |
| | XX | XXX.X | XX |
| | XX | XXX.X | XX |

%=(n/N)\*100

Dose Reduction: at cycle start


[Program Path; Date/Time Produced; Date Data Extract].

#### Programming Notes:

Patients are to be counted just once per tr. modification category. Cycles at which multiple occurrences of the same tr. modification category were reported are to be counted just once per tr. modification category.

Appendix 2.3.6 – Treatment Exposure: Frequency Distributions of Patients by Reasons for Treatment Modifications - Treated Patients –

Page by Regimen

| Treated Patients (N=xx) | No. of Patients | |
|------------------------------------|-----------------|-------|
| Reasons for Treatment Modification | n | % |
| Any Reason | XX | XXX.X |
| | XX | XXX.X |
| | XX | XXX.X |
| Hematological toxicity | XX | XXX.X |
| | XX | XXX.X |
| | XX | XXX.X |
| Non-hematological toxicity | XX | XXX.X |
| | XX | XXX.X |
| | XX | XXX.X |
| Other | XX | XXX.X |
| | XX | XXX.X |
| | XX | XXX.X |
| Unknown Reason | XX | XXX.X |
| | XX | XXX.X |
| | XX | XXX.X |

%=(n/N)\*100


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

n: count patients for each toxicity class (i.e. hematological/non-hematological/other), regardless of what kind of treatment modification is performed; if multiple occurrences of the same toxicity class are reported within a cycle or throughout different cycles patients are to be counted just once per class.

#### Appendix 2 – Section 4 – Treatment Efficacy

Appendix 2.4.1.<x> – Treatment Efficacy: Progression Free Survival Rate at 3 Months
- Evaluable Patients/Treated –

Page by Regimen

| Progression Free Survival at 3 Months | Evaluable Patients/ Treated (N=xx) | | | |
|---|---|---|---|---|
| | n | % | 95 % CI - LL | 95 % CI - UL |
| Success | XX | XXX.X | XX.XX | XX.XX |
| Failure | XX | XXX.X | | |
| Total | XX | XXX.X | | |

%=(n/N)\*100. N=no. of treated/evaluable patients

Success: Patients who were progression free for longer than 91 days (i.e. 3 months) and with an overall response at the 3rd month assessment equal to SD or better. Valid assessments were to be within day 134; the outcome of assessments performed outside this time window was considered as failure regardless of the outcome recorded.

Failure: All patients who were not success. 95% CI: Exact Binomial Confidence Limits


Figure 2.4.1.<x> – Treatment Efficacy: Kaplan-Meier Curve for Progression Free Survival - Evaluable Patients/Treated –

Page by Regimen

Progression Free Survival (months): from the treatment start date to the date of death from any cause Median Progression Free Survival (95% CI): xx.xx (xx.xx - xx.xx)


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Create three versions of the graph: the graph automatically created by the SAS proc lifetest - Kaplan-Meier method ( .gif format) as control, and two other graphs obtained by plotting the relevant variables with SAS proc gplot (same procedure, two different output file formats: .gif and .pdf )

"General Footnotes" not to be printed for .gif graphs.

Appendix 2.4.2.<x> - Treatment Efficacy: Best Confirmed Tumor Response - Evaluable/Treated -

# Page by Regimen

| | Treated / Evaluable Patients | | | |
|---|---|---|---|---|
| Best Confirmed Tumor Response | (N=xx) | | | |
| | n | % | 95 % CI - LL | 95 % CI - UL |
| Objective Response (CR + PR) | XX | XXX.X | XXX.XX | XXX.XX |
| Disease Control (CR+PR+SD) | XX | XXX.X | XXX.XX | XXX.XX |
| Complete Response (CR) | XX | XXX.X | | |
| Partial Response (PR) | XX | XXX.X | | |
| Progression of Disease (PD) | XX | XXX.X | | |
| Not Evaluable | XX | XXX.X | | |

%=(n/N)\*100. N=no. of treated patients. 95% CI: Exact Binomial Confidence Limits


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

95% CI: 95% Exact Confidence Limits for tumor response rate.

Valid Response values CR, PR, SD, PD, NE

Appendix 2.4.3.<x> – Treatment Efficacy: Best Unconfirmed Tumor Response - Evaluable/Treated -

Page by Regimen

| Best Unconfirmed Tumor Response | Treated / Evaluable Patients (N=xx) | |
|---|---|---|
| | n | % |
| Overall Response (CR + PR) | XX | XXX.X |
| Complete Response (CR) | XX | XXX.X |
| Partial Response (PR) | XX | XXX.X |
| Stable Disease (SD) | XX | XXX.X |
| Progression of Disease (PD) | XX | XXX.X |
| Not Evaluable (NE) | XX | XXX.X |

Unconfirmed Tumor Response: for each patient it's the best response reported throughout the study period as overall response, regardless of the confirmation.

%=(n/N)\*100. N=no. of treated patients.


[Program Path; Date/Time Produced; Date Data Extract]

Programming Notes:

Valid Response values CR, PR, SD,PD, NE
Appendix 2.4.4.<x> – Treatment Efficacy: Statistical Analysis of Time-To-Event Endpoints – Treated / Evaluable Patients –

### Page by Regimen

| Treated / Evaluable Patients (N=xx) | No. of<br>Pts. | No. of<br>Events | Min | Max | Median | Median 95% CI -<br>LL | Median 95% CI - UL |
|---|---|---|---|---|---|---|---|
| Progression Free Survival (months) | XX | XX | XXX.XX | xxx.xx + | XXX.XX | XXX.XX | XXX.XX |
| Overall Survival (months) | XX | XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Duration of response (months) | XX | XX | XXX.XX | xxx.xx + | XXX.XX | XXX.XX | XXX.XX |

N=: no. of treated (evaluable) patients.

No. of Events: the no. of failure patients for the given endpoint.

Median: estimated by the Kaplan-Meier method.

+: Censored observation

Overall survival: from the treatment start date to the date of death from any cause

Progression free survival: from the treatment start date to the date of objective progression or death from any cause

Duration of response: from the date when response was first assessed to the date of progression or date of censoring, whichever comes first


[Program Path; Date/Time Produced; Date Data Extract]

# **Programming Notes:**

Summary statistics are to be calculated by SAS PROC LIFETEST using the Kaplan-Meier method.

Figure 1.9.2.<x> – Treatment Efficacy: Kaplan-Meier Curve for Overall Survival - Treated / Evaluable Patients—

Page by Regimen

Median Progression Free Survival (95% CI): xx.xx (xx.xx - xx.xx)


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Create three versions of the graph: the graph automatically created by the SAS proc lifetest - Kaplan-Meier method ( .gif format) as control, and two other graphs obtained by plotting the relevant variables with SAS proc gplot (same procedure, two different output file formats: .gif and .pdf)

"General Footnotes" not to be printed for .gif graphs.

Appendix 2.4.5 – Treatment Efficacy: ECOG Performance Status: On Treatment Worst Assessment vs. Pretreatment - Treated Patients with at Least One Assessment On Treatment -

# Page by Regimen

| Treated Patients (N=xx) | | On-Treatment Worst Assessment | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | 0 | | 1 | ٠ | | Тс | otal |
| Pretreatment Assessment | n | % | n | % | n | % | n | % |
| Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| 2 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| >2 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Unknown | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100.

N = treated patients with at least one Performance Status assessment after treatment start date.


[Program Path; Date/Time Produced; Date Data Extract]

# Appendix 2 – Section 5 – Adverse Events

Appendix 2.5.1 – Adverse Events: Patients with on Treatment AEs by System Organ Class and Maximum CTC Grade - Treated Patients –

#### Page by Regimen

| Treated Patients (N=xx) | | Maximum CTC Grade | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| , , , | Any ( | Any Grade 3-4 1 Unk | | | | | | | | |
| System Organ Class | n | % | n | % | n | % | n | % | n | % |
| Any System | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC 1] | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC n] | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

# **Programming Notes:**

Within each "by group", sort SOCs by descending frequency of "Any Grade"

For each SOC (System Organ Class), count patients according to the maximum CTC grade reported for that SOC.

Appendix 2.5.2 – Adverse Events: Patients with on Treatment AEs by AE MedDRA Preferred Term and Maximum CTC Grade - Treated Patients –

# Page by Regimen

| Treated Patients (N=xx) | | Maximum CTC Grade | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treated rationts (TV XX) | Any Grade 3-4 1 | | | | | | | U | nk | |
| Preferred Term | n | % | n | % | n | % | n | % | n | % |
| Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [Term 1] | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [Term i] | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Within each "by group", sort AEs by descending frequency of "Any Grade".

For each AE (i.e. for each Preferred Term), count patients according to the maximum CTC grade reported for that event.

Appendix 2.5.3 – Adverse Events: Patients with on Treatment AEs by SOC, AE MedDRA Preferred Term and Maximum CTC Grade - Treated Patients -

# Page by Regimen

| Trantad Dati | anta (N-vv) | | | | Ma | aximum | CTC Gra | ade | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treated Pati | ents (N-xx) | Any | Grade | 3 | -4 | | 1 | | ••• | U | nk |
| System Organ Class | Preferred Term | n | % | n | % | n | % | n | % | n | % |
| Any System | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | xxx.x |
| [SOC 1] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event i | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | ••• | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC i] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

### **Programming Notes:**

Within each by group, SOC and AE (i.e. for each Preferred Term), count patients according to the maximum CTC grade reported for that event and sort SOCs by descending frequency of "Any Term" at "Any Grade".

Appendix 2.5.4 – Adverse Events: Patients with AEs with Possible to Definite Relationship to Study Treatment by SOC and Maximum CTC Grade

- Treated Patients –

# Page by Regimen

| Treated Patients (N=xx) | | Maximum CTC Grade | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Ar | ıy Grade | 3 | -4 | | 1 | | •• | Uı | ık |
| System Organ Class | n | % | n | % | n | % | n | % | n | % |
| Any System | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC 1] | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC n] | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

# **Programming Notes:**

Within each "by group", sort SOCs by descending frequency of "Any Grade".

For each SOC (System Organ Class), count patients according to the maximum CTC grade reported for that SOC.

Appendix 2.5.5 – Adverse Events: Patients with AEs with Possible to Definite Relationship to Study Treatment by AE MedDRA Preferred Term and Maximum CTC Grade

- Treated Patients –

# Page by Regimen

| Treated Patients (N=xx) | | Maximum CTC Grade | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treated ratients (N=XX) | Any | Grade | 3 | 3-4 | | 1 | | | | Unk |
| Preferred Term | n | % | n | % | n | % | n | % | n | % |
| Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [Term 1] | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [Term i] | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | | | | | | • • • | | |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Within each "by group", sort AEs by descending frequency of "Any Grade"

For each AE (i.e. for each Preferred Term), count patients according to the maximum CTC grade reported for that event.

Appendix 2.5.6 – Adverse Events: Patients with AEs with Possible to Definite Relationship to Study Treatment by SOC, AE MedDRA Preferred Term and Maximum CTC Grade

- Treated Patients –

#### Page by Regimen

| Tracted Detion | ota (N-vv) | | | | Max | imum ( | CTC Gra | de | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treated Patier | its (IV=XX) | Any | Grade | | 3-4 | | 1 | | | | Unk |
| System Organ Class | Preferred Term | n | % | n | % | n | % | n | % | n | % |
| Any System | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC 1] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event i | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC i] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Within each "by group", SOC and AE (i.e. for each Preferred Term), count patients according to the maximum CTC grade reported for that event and sort SOCs by descending frequency of "Any Term" at "Any Grade".

Appendix 2.5.7 – Adverse Events: Patients with on Treatment Serious AEs by SOC, AE MedDRA Preferred Term and Maximum CTC Grade - Treated Patients –

# Page by Regimen

| Trantad Do | tionta (N-vv) | | | | Max | imum ( | CTC Gra | de | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treateu Fa | tients (N=xx) | Any | Grade | | 3-4 | | 1 | | • • • | | Unk |
| System Organ Class | Preferred Term | n | % | n | % | n | % | n | % | n | % |
| Any System | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC 1] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event i | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC i] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

### **Programming Notes:**

Within each "by group", SOC and AE (i.e. for each Preferred Term), count patients according to the maximum CTC grade reported for that event and sort SOCs by descending frequency of "Any Term" at "Any Grade".

Appendix 2.5.8 – Adverse Events: Patients with Serious AEs with Possible to Definite Relationship to Study Treatment by SOC, AE MedDRA Preferred Term and Maximum CTC Grade

- Treated Patients –

# Page by Regimen

| Trantad De | atients (N=xx) | | | | Max | imum ( | CTC Gra | de | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treated Fa | atients (N-xx) | Any | Grade | | 3-4 | | 1 | | ••• | | Unk |
| System Organ Class | Preferred Term | n | % | n | % | n | % | n | % | n | % |
| Any System | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC 1] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event i | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | ••• | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC i] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | ••• | | | | | | | | | | |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Within each "by group", SOC and AE (i.e. for each Preferred Term), count patients according to the maximum CTC grade reported for that event and sort SOCs by descending frequency of "Any Term" at "Any Grade".

Appendix 2.5.9 – Adverse Events: Patients with on Treatment AEs Leading to Withdrawal from Study Treatment by SOC, AE MedDRA Preferred Term and Maximum CTC Grade

- Treated Patients –

# Page by Regimen

| Tracted Dati | onto (N-vv) | | | | Max | imum C | TC Gra | de | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treated Pati | ents (N-XX) | Any | Grade | 3 | -4 | | 1 | | | J | J <b>nk</b> |
| System Organ Class | Preferred Term | n | % | n | % | n | % | n | % | n | % |
| Any System | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC 1] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Event i | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| [SOC i] | Any Term | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

Only AEs whose Action Taken was "Drug Permanently Withdrawn" are displayed.

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Select AE with action taken=drug permanently withdrawn.

Within each by group, SOC and AE (i.e. for each Preferred Term), count patients according to the maximum CTC grade reported for that event and sort SOCs by descending frequency of "Any Term" at "Any Grade"

Appendix 2.5.10 – Deaths: Frequency of Death according to Most Probable Cause and Time of Occurence - Treated Patients –

Page by Regimen

| Treated Patients (N=xx) | , | Total | Treatr | Days since<br>nent Last<br>Dose | Treat | Days since<br>tment Last<br>Dose |
|---|---|---|---|---|---|---|
| Most Probable Cause | n | % | n | % | n | % |
| Any cause | XX | XX.X | XX | XX.X | XX | XX.X |
| Progressive Disease | XX | XX.X | XX | XX.X | XX | XX.X |
| Adverse Event | XX | XX.X | XX | XX.X | XX | XX.X |
| | | ••• | • • • | | | ••• |
| Unknown | XX | XX.X | XX | XX.X | XX | XX.X |

%=(n/N)\*100

N = no. of treated patients


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

See ADP for classification of causes of death vs source of info.

# Appendix 2 - Section 6 - Laboratory Assessments

Appendix 2.6.1 – Hematology: Frequency Distribution of Patients based on Maximum CTC Grade On Treatment versus Pretreatment

- Treated Patients with at Least One Assessment On Treatment 
- All Cycles, Cycle 1, Cycles > 1-

Page by Regimen / Laboratory Test: < WBC >

| | | | Maximum CTC Grade on Treatment | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | ( | ) | | | 4 | | To | otal |
| Study Period | | Pretreatment CTC Grade | n | % | n | % | n | % | n | % |
| All Cycles | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | • | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Unknown | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle 1 | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle >1 | (N=xx) | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

N = treated patients with at least one assessment after treatment start date.

%=(n/N)\*100.

Only lab. tests included in the NCI CTCAE v3.0 document. Maximum CTC Grade: the Maximum CTC grade reported for each treated patient and each lab test during the treatment period.


[Program Path; Date/Time Produced; Date Data Extract]

Programming Notes:

Sort by "page by variables".

Appendix 2.6.2 – Hematology: Frequency Distribution of Treatment Cycles based on Maximum CTC Grade On Treatment versus Pretreatment - Cycles with at Least One Assessment - All Cycles, Cycle 1, Cycles > 1 -

Page by Regimen / Laboratory Test: < WBC >

| | | | | Ma | ximum | CTC G | rade or | Treatm | ent | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | ( | 0 | | | | 4 | Total | |
| Study Period | | Pretreatment CTC<br>Grade | n | % | n | % | n | % | n | % |
| All Cycles | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Unknown | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle 1 | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle >1 | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | •••• | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

N =cycles with at least one assessment

%=(n/N)\*100.

Only lab. tests included in the NCI CTCAE v3.0 document. Maximum CTC Grade: the Maximum CTC grade reported for each cycle and each lab test during the treatment period.


[Program Path; Date/Time Produced; Date Data Extract]

<u>Programming Notes</u>:

Sort by "page by variables".

Appendix 2.6.3 – Blood Chemistry: Frequency Distribution of Patients based on Maximum CTC Grade On Treatment versus Pretreatment (Part I)

- Treated Patients with at Least One Assessment On Treatment 
- All Cycles, Cycle 1, Cycles > 1-

Page by Regimen / Laboratory Test: < AST >

| | | | | Ma | ximum | CTC G | rade or | Treatm | ent | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 0 | | | 4 | | To | otal |
| Study Period | | Pretreatment CTC | n | % | n | % | n | % | n | % |
| | | Grade | | | | | | | | |
| All Cycles | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle 1 | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle >1 | (N=xx) | Total | XX | xxx.x | XX | XXX.X | XX | xxx.x | XX | xxx.x |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | •••• | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

N = treated patients with at least one assessment after treatment start date.

%=(n/N)\*100.

(Part I): Only lab. tests included in the NCI CTCAE v3.0 document and whose abnormality is determined by one-way modifications only.

Maximum CTC Grade: the Maximum CTC grade reported for each treated patient and each lab test during the treatment period.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by "page by variables".

Appendix 2.6.4 – Blood Chemistry: Frequency Distribution of Patients based on Maximum CTC Grade On Treatment versus Pretreatment (Part II)

- Treated Patients with at Least One Assessment On Treatment -

- All Cycles -

Page by Regimen / Laboratory Test: < Sodium >

| | | | <h< th=""><th>yper/ Hy</th><th>/po&gt; - N</th><th><b>Maximun</b></th><th>n CTC (</th><th>Grade on</th><th>Treatm</th><th>ent</th></h<> | yper/ Hy | /po> - N | <b>Maximun</b> | n CTC ( | Grade on | Treatm | ent |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | 1 | | | | 5 | | To | tal |
| Study Period | | Pretreatment CTC Grade | n | % | n | % | n | % | n | % |
| All Cycles | (N=xx) | Total | XX | XX.X | XX | XX.X | XX | XX.X | XX | XX.X |
| | | 4 (H) | | | | | | | | |
| | | 3 (H) | | | XX | XX.X | XX | XX.X | XX | XX.X |
| | | 2 (H) | | | | | | | | |
| | | 1 (H) | | | | | | | | |
| | | 0 | | | | | | | | |
| | | 1 (L) | | | | | | | | |
| | | 2 (L) | | | | | | | | |
| | | 3 (L) | | | | | | | | |
| | | 4 (L) | | | | | | | | |
| | | Not Assessed | | | | | | | | |

N = treated patients with at least one assessment after treatment start date.

%=(n/N)\*100.

(Part II): Only lab. tests included in the NCI CTCAE v3.0 document and whose abnormality is determined by two-way modifications.

Maximum CTC Grade: the Maximum treatment emergent CTC grade reported for each treated patient during the treatment period.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by "page by variables".

Select collected lab tests listed in NCI CTCAE v3.0 for which both 'hyper' and 'hypo' grading is provided. For this study: Magnesium, Potassium, Sodium.

Appendix 2.6.5 – Blood Chemistry: Frequency Distribution of Treatment Cycles based on Maximum CTC Grade On Treatment versus Pretreatment (Part I)

- Cycles with at Least One Assessment 
- All Cycles, Cycle 1, Cycles > 1 -

Page by Regimen / Laboratory Test: < AST >

| | | | | Ma | ximum | CTC G | rade or | Treatm | ent | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 0 | | | 4 | | To | otal |
| Study Period | | Pretreatment CTC | n | % | n | % | n | % | n | % |
| | | Grade | | | | | | | | |
| All Cycles | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Unknown | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle 1 | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle >1 | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

N =cycles with at least one assessment.

%=(n/N)\*100.

(Part I): Only lab. tests included in the NCI CTCAE v3.0 document and whose abnormality is determined by one-way modifications only.

Maximum CTC Grade: the Maximum CTC grade reported for each cycle and each lab test during the treatment period.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by "page by variables".

Appendix 2.6.6 – Blood Chemistry: Frequency Distribution of Treatment Cycles based on Maximum CTC Grade On Treatment versus Pretreatment (Part II)

- Cycles with at Least One Assessment 
- All Cycles-

Page by Regimen / Laboratory Test: < Sodium >

| | | | <hyper hypo=""> - Maximum CTC Grade</hyper> | | | | | Grade on | n Treatment | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 1 | | | 5 | | To | otal |
| Study Period | | Pretreatment CTC Grade | n | % | n | % | n | % | n | % |
| All Cycles | (N=xx) | Total | XX | XX.X | XX | XX.X | XX | XX.X | XX | XX.X |
| | | 4 (H) | | | | | | | | |
| | | 3 (H) | | | XX | XX.X | XX | XX.X | XX | XX.X |
| | | 2 (H) | | | | | | | | |
| | | 1 (H) | | | | | | | | |
| | | 0 | | | | | | | | |
| | | 1 (L) | | | | | | | | |
| | | 2 (L) | | | | | | | | |
| | | 3 (L) | | | | | | | | |
| | | 4 (L) | | | | | | | | |
| | | Not Assessed | | | | | | | | |

N = cycles with at least one assessment.

%=(n/N)\*100.

(Part II): Only lab. tests included in the NCI CTCAE v3.0 document and whose abnormality is determined by two-way modifications.

Maximum CTC Grade: the Maximum treatment emergent CTC grade reported for each cycle and each lab test during the treatment period.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by "page by variables".

Select collected lab tests listed in NCI CTCAE v3.0 for which both 'hyper' and 'hypo' grading is provided. For this study: Magnesium, Potassium, Sodium

Appendix 2.6.7 – Coagulation: Frequency Distribution of Patients based on Maximum CTC Grade On Treatment versus Pretreatment - Treated Patients with at Least One Assessment On Treatment - All Cycles, Cycle 1, Cycles > 1 –

Page by Regimen / Laboratory Test: < INR >

| Study P | laria d | | | Ma | ximum | CTC G | rade or | 1 Treatm | ent | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study P | erioa | | | 0 | | •• | | 4 | Т | otal |
| | | Pretreatment CTC<br>Grade | n | % | n | % | n | % | n | % |
| All Cycles | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | •••• | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Unknown | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle 1 | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | · | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle >1 | (N=xx) | 0 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | 1 | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

N = treated patients with at least one assessment after treatment start date %=(n/N)\*100.

Only lab. tests included in the NCI CTCAE v3.0 document. Maximum CTC Grade: the Maximum CTC grade reported for each treated patient and each lab test during the treatment period.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by "page by variables".

Appendix 2.6.8 – Laboratory Tests without a NCI-CTC Grade: Frequency Distribution of Patients Based on On Treatment Worst Assessment versus Pretreatment - Treated Patients with at Least One Assessment On Treatment - All Cycles, Cycle 1, Cycles > 1 –

Page by Regimen - <Panel>: e.g. Hematology Laboratory Test: < Eosinophils >

| | | | | On Treati | ment Worst A | ssessmen | nt | | |
|---|---|---|---|---|---|---|---|---|---|
| Study Period | | Above | e UNL | With | nin NLs | Belo | w LNL | To | otal |
| | Pretreatment Value | n | % | n | % | n | % | n | % |
| All Cycles (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Above ULN | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Within NLs | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Below LLN | XX | XXX.X | XX | XXX.X | XX | XXX.X | | |
| | Not Assessed | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Cycle 1 (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | Above ULN | XX | XXX.X | XX | XXX.X | XX | XXX.X | | |
| | Within NLs | XX | XXX.X | XX | XXX.X | XX | XXX.X | | |
| | Below LLN | XX | XXX.X | XX | XXX.X | XX | XXX.X | | |
| | Not Assessed | | | | | | | | |
| Cycle >1 (N=xx) | | XX | XXX.X | XX | XXX.X | XX | XXX.X | | |
| | | XX | XXX.X | XX | XXX.X | XX | XXX.X | | |

N = treated patients with at least one assessment after treatment start date %=(n/N)\*100.


[Program Path; Date/Time Produced; Date Data Extract]

### **Programming Notes:**

Sort by "page by variables".

Blood Chemistry - < Lab Test >: Blood Urea Nitrogen (BUN), Urea (Carbamide) Blood, Chloride.

# Appendix 2.7 – Other Safety Assessments

Appendix 2.7.1 – Other Safety Assessments: Blood Pressure - On Treatment Worst Assessment versus Pretreatment - Treated Patients with at Least One Assessment On Treatment -

Page by Regimen

| Tracted Datients (N-vv) | | On-Treatment Worst Assessment | | | | |
|---|---|---|---|---|---|---|
| Treated Patients (N=xx) | No | Normal | | ormal | Тс | otal |
| Pretreatment Assessment | n | % | n | % | n | % |
| Total | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Normal | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Abnormal | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Unknown | XX | XXX.X | XX | XXX.X | XX | XXX.X |

Normal: systolic blood pressure < 140 and diastolic blood pressure < 90 Abnormal: systolic blood pressure  $\ge 140$  or diastolic blood pressure  $\ge 90$ .

%=(n/N) \* 100. N = treated patients with at least one blood pressure measurement after treatment start date.


[Program Path; Date/Time Produced; Date Data Extract]

Appendix 2.7.2 – Other Safety Assessments: ECG - On Treatment Assessment versus Pretreatment Condition - Treated Patients with at Least One Assessments On Treatment -

Page by Regimen

| Tracted Detients (N-vv) | On-Treatment ECG Abnormality | | | | | |
|---|---|---|---|---|---|---|
| Treated Patients (N=xx) | N | О | At leas | t One | Total n % xx xx.2 xx xx.2 xx xx.2 | otal |
| Pretreatment ECG Abnormality | n | % | n | % | n | % |
| Total | XX | XX.X | XX | XX.X | XX | XX.X |
| No | XX | XX.X | XX | XX.X | XX | XX.X |
| Yes | XX | XX.X | XX | XX.X | XX | XX.X |
| Unknown | XX | XX.X | XX | XX.X | XX | XX.X |

%=(n/N)\*100.

N = treated patients with at least one EGC assessment after treatment start date.


[Program Path; Date/Time Produced; Date Data Extract]

Appendix 2.7.3 – Other Safety Assessments: ECG - On Treatment Abnormality Findings - Treated Patients with at Least One Assessment On Treatment –

Page by Regimen

| Abnormality Category | Treated P | atients (N=xx) |
|----------------------|-----------|----------------|
| Abhormanty Category | n | % |
| Rhythm | XX | XXX.X |
| P-Wave Morphology | XX | XXX.X |
| Conduction | XX | XXX.X |
| QRS | XX | XXX.X |
| ST-T Wave | XX | XXX.X |
| | XX | XXX.X |

%=(n/N)\*100.

N = treated patients with at least one EGC assessment after treatment start date.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Abnormality categories: count patients within each category. If multiple occurrences of the same abnormality (e.g. conduction) are reported, the patient should be counted only once.

Appendix 2.7.4 – Other Safety Assessments: Funduscopic Examination - On Treatment Worst Assessment versus Pretreatment - Treated Patients with at Least One Assessment On Treatment -

# Page by Regimen

| | | | | | | On-Treatment Wor | st Assessment | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | No | rmal | Abnormal, not o | clinically relevant | Abnormal, cl | linically relevant | Te | otal |
| Fundus | | Pretreatment Assessment | n | % | n | % | n | % | n | % |
| Right Eye | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Normal | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Abnormal, not clinically relevant | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Abnormal, clinically relevant | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Unknown | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| Leftt Eye | (N=xx) | Total | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Normal | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Abnormal, not clinically relevant | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Abnormal, clinically relevant | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |
| | | Unknown | XX | XXX.X | XX | XXX.X | XX | XXX.X | XX | XXX.X |

%=(n/N)\*100.

N = treated patients with at least one assessment after treatment start date.

[Protocol No.; Study Description] [Program Path; Date/Time Produced; Date Data Extract]

APPENDIX 3: INDIVIDUAL DATA LISTINGS

# Appendix 3 - Section 1 - Patient Disposition

Appendix 3.1.1 – Patient Disposition: Patient Registration – Registered Patients –

| Enrolled<br>Pt | Treated<br>Pt | Pt.<br>No. | Pt.<br>Screening<br>No. | Center No. | Age<br>/Sex<br>/Race | Date of Birth | Date of Informed<br>Consent | Date of<br>Enrollment |
|---|---|---|---|---|---|---|---|---|
| N | N | Sxxx | | XXXXX | 35/M/W | ddmmmyyyy | ddmmmyyyy | |
| N | N | Sxxx | | XXXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | |
| Y | N | XXXX | Sxxx | XXXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy |
| Y | Y | XXXX | Sxxx | XXXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy |
| Y | Y | XXXX | Sxxx | XXXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy |
| Y | Y | XXXX | Sxxx | XXXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy |

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.


[Program Path; Date/Time Produced; Date Data Extract]

# <u>Programming Notes:</u>

Sort by enrolled patients (N, Y), treated patients (N, Y), patient no.

Pt. Screening No.: for enrolled patients it is reported on the patient enrollment page of CRF.

Date of informed consent: it is reported on the demography page of CRF.

Appendix 3.1.2 – Patient Disposition: Registered but Not Enrolled Patients - Screening Failures -

| Pt. No. | Center<br>No. | Date of Informed<br>Consent | Reason for Screening Failure | Other Reason, specify | Comments |
|---|---|---|---|---|---|
| Sxxx | XXXXX | ddmmmyy | Inclusion/Exclusion Criteria not fulfilled | | _ |
| Sxxx | XXXXX | ddmmmyy | Other: | | |
| Sxxxx | XXXXX | ddmmmyy | | | |
| Sxxxx | XXXXX | ddmmmyy | | | |
| Sxxxx | XXXXX | ddmmmyy | | | |


[Program Path; Date/Time Produced; Date Data Extract]

# **Programming Notes:**

Sort by patient no.

Reason for Screening Failure: it is reported on the screening failure page of CRF

# Appendix 3.1.3 – Patient Disposition: Summary of Patient Information - Enrolled Patients-

### Page by Regimen

| Pt. No | First Dose<br>Date | Last Dose<br>Date | Cum. Dose<br>(mg | Total<br>No. of<br>Cycles | Tr.<br>Status | Time on<br>Treat.<br>(weeks) | Primary<br>Off Tr.<br>Reason | End of AE<br>Reporting<br>Period | FU<br>Status | Study<br>Status | Last<br>Recorded<br>Date | | Time on<br>Study<br>( weeks ) | Primary Off Study<br>Reason |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | ddmmmyy | ddmmmyy | XXX.X | 1 | Off. | XXX.X | AE | ddmmmy | On FU | On | ddmmmyy | | XX | XXXXXXXX |
| XXXX | ddmmmyy | ddmmmyy | XXX.X | 4 | | XXX.X | Pt's refusal | | No FU | Off | ddmmmyy | § | XX | XXXXXXXX |
| XXXX | ddmmmyy | ddmmmyy | XXX.X | 2 | Off | XXX.X | Progression | ddmmmy | - | Off | ddmmmyy | | XX | XXX XXXXX |

Time on Treatment: time from the first dose date to last dose date

Time on Study: time from the informed consent date to the last recorded date

(§) Last Recorded Date is different from Investigator's Decision date or Consent Withdrawn date in the Off Study form


[Program Path; Date/Time Produced; Date Data Extract]

Programming Notes:

Sort by patient no.

Cumulative dose: from start to end of treatment.

Usually Time Unit of Time on Study is the same as for Duration of Treatment, but it is not mandatory, i.e. could be weeks and months respectively.

# Appendix 3.1.4 – Patient's Survival Status during Follow Up - Treated Patients-

# Page by Regimen

| Pt. No | Visit | Status | Alive as of:<br>Date | Last Known<br>Alive Date | Date of<br>Death | Most<br>Probable<br>Cause | Details |
|---|---|---|---|---|---|---|---|
| XXXX | FU-1 | Alive | ddmmmyyyy | | | | |
| | | •••• | | | | D | |
| | FU-2 | Expired | | | ddmmmyyyy | Progressive<br>Disease | XXXXXXXXXXX |
| XXXX | FU-1 | Lost to FU | ••• | ddmmmyyyy | ••• | | |


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by patient no., visit

By regimen: in this study one regimen only: 150 mg/day x 7 days q 2 wks

# Appendix 3 - Section 2 - Protocol Deviations

Appendix 3.2.1 - Protocol Deviations: Violations of Inclusion / Exclusion Criteria - Enrolled Patients -

#### Page by Regimen

| Treated | Pt. | Center | Criterion | Criterion | Y/N | |
|---------|------|--------|-----------|-----------|--------|---|
| Pt. | No. | No. | Number | Chenon | 1 / 1N | |
| N | XXXX | XXXX | IC01 | | Y | |
| | | | IC02 | | N | * |
| | | | EC01 | | Y | * |
| | | | EC02 | | N | |
| | | | • • • • | •••• | | |
| Y | XXXX | XXXX | IC01 | •••• | N | * |

Only patients with at least one protocol deviation and/or waiver granted are displayed. The \* identified the protocol deviation. IC: Inclusion Criterion; EC: Exclusion Criterion


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by treated patients (N, Y), patient no, Criterion no. (incl., excl.).

Only patients with at least one protocol deviation or missing evaluation and/or waiver granted are to be displayed

# Appendix 3 – Section 3 – Patients Evaluability for Efficacy Analysis

Appendix 3.3.1 –Evaluability for Efficacy Analysis: Evaluability Criteria and Individual Evaluability Status - Enrolled Patients-

| | Dose Cy1+Cy2 | Tumor Assessment | | | | |
|---|---|---|---|---|---|---|
| Pt. No | >/= 80% cum. intended dose | at Pretreat. | On<br>Treat. | Death Before 1st<br>Tumor Assessment | Eval.Pt. | Reasons for<br>Non-<br>Evaluability |
| XXXX | Y | Y | Y | N | Y | |
| XXXX | Y | Y | Y | Y | Y | |
| XXXX | N | Y | Y | | N | R1 |
| XXXX | XX.X | N | Y | N | N | R3 |
| XXXX | XX.X | N | N | N | N | R4 |
| XXXX | N | Y | Y | N | N | R2 |
| XXXX | XX.X | Y | N | Y | Y | |
| XXXX | XX.X | Y | Y | N | N | R3 |

#### Reasons for Non-Evaluability:

R1: the patient didn't receive at least 80% of the intended dose for the first two treatment cycles

R2: the pretreatment oncologic assessment was not performed

R3: no on treatment oncologic assessment was performed and the patient didn't die before the first scheduled (re)assessment

## [Protocol No. (Study Description)]

[program path; date/time produced; date data extract]

#### Programming notes:

Sort by patient no.

# Appendix 3 – Section 4 – Demography and Pretreatment

Appendix 3.4.1 - Demography and Pretreatment: Tumor History - Primary Diagnosis - Treated Patients -

#### Page by Regimen

| Pt.<br>No | Age<br>/Sex<br>/Race | Primary Diagnosis | Type of Diagnosis | Date of<br>Diagnosis | Months to<br>Tr. Start | | WHO<br>Classification | Masaoka<br>Stage |
|---|---|---|---|---|---|---|---|---|
| XXXX | 38/M/W<br>xx/x/x | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Cytological<br>Histological | ddmmmyyyy<br>mmmyyyy | XXX.X<br>XXX.X | * | B3<br>C | II<br>IIB |
| XXXX | | | | | | | ••• | |
| XXXX | | | ••• | ••• | ••• | | | UNK |
| XXXX | | | | ••• | | | | |

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.

B3= Well-differentiated thymic carcinoma, C= Tymic Carcinoma

Months to Tr. Start: From date of primary diagnosis to treatment start date.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by pt no.

<sup>\*:</sup> Estimated time when incomplete date was reported.

# Appendix 3.4.2 - Demography and Pretreatment: Tumor History – Diagnosis at Study Entry - Treated Patients –

#### Page by Regimen

| Pt.<br>No | Age/Sex<br>/Race | Extent at<br>Study Entry | Date of<br>Current<br>Diagnosis | Weeks to<br>Tr. Start | Masaoka<br>Stage | Total No. of Recurrences /Progression | Sites of<br>Metastatic<br>Disease | Specify | Months from Primary Diagnosis |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | 38/M/W | Locally | ddmmmyyyy | XXX.X | II | 1 | | | xxx.x * |
| xxxx | xx/x/xx | Advanced<br>Metastatic | уууу | xxx.x * | IIB<br> | 3 | Lung<br>Bone | | xxx.x * |
| xxxx | xx/x/xx | Metastatic | ddmmmyyyy | XXX.X | | X | Brain Lymph nodes Other | xxxxxxxxxxx | xxx.x |

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.

Weeks to Tr. Start: From date of diagnosis to treatment start date.

Total No. of Recurrences /Progression: including current one.

Months from Primary Diagnosis: From initial diagnosis date to current diagnosis date.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by pt no.

<sup>\*:</sup> Estimated time when incomplete date was reported.

Appendix 3.4.3 - Demography and Pretreatment: Tumor History – NCI Confirmation of Diagnosis - Treated Patients –

# Page by Regimen

| Pt.<br>No. | WHO<br>Classification<br>by Investigator | Date of<br>Diagnosis by<br>Institution | Tumor Type at Diagnosis according to Institution | Thymic Carcinoma<br>Type Confirmed by<br>Institution? | Details of Thymi<br>Carcinoma (C) | Details of Thymic Carcinoma (C), Specify | Other Tumor<br>Type, Specify | Comments |
|---|---|---|---|---|---|---|---|---|
| XXXX | В3 | ddmmmyyyy | В3 | Y | | | | |
| XXXX | C | ddmmmyyyy | Other | N | * | | XXXXXXXX | |
| XXXX | C | ddmmmyyyy | C | Y | Other | xxxxxxxx | | |
| XXXX | C | ddmmmyyyy | Other | | * | | XXXXXXXX | XXXXXXXX |

B3= Well-differentiated thymic carcinoma, C= Thymic Carcinoma Tumor Type at Diagnosis by Independent Reviewer: \* if Other


[Program Path; Date/Time Produced; Date Data Extract]

# <u>Programming Notes</u>:

Sort by pt no., date of diagnosis by independent reviewer.

# Appendix 3.4.4 - Demography and Pretreatment: History of Other Cancers - Treated Patients—

### Page by Regimen

| Pt. No | Agg/Coy/Dogg | Site of | Histological | Date of | Months to | |
|---|---|---|---|---|---|---|
| | Pt. NO | Age/Sex/Race | Tumor | Type | Diagnosis | Tr. Start |
| | XXXX | 38/M/W | XXXXXXX | XXXXXXX | ddmmmyyyy | XXX.X |
| | XXXX | xx/x/xx | XXXXXXX | XXXXXXX | уууу | xxx.x * |
| | XXXX | xx/x/xx | XXXXXXXX | XXXXXXXX | ddmmmyyyy | XXX.X |

Only patients with at least one other cancer are displayed.

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.

Months to Tr. Start: From date of diagnosis of other cancer to treatment start date.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by pt no., line no. (no print).

Select only patients with Other Cancer = 'yes' or derived 'yes'.

<sup>\*:</sup> Estimated time when incomplete date was reported.
## Appendix 3.4.5 - Demography and Pretreatment: Tumor History - Prior Antitumor Treatments/Procedures - Treated Patients -

### Page by Regimen

| Pt. No | Primary<br>Diagnosis | Chron.<br>Seq. No. | Start Date | Stop Date | Weeks to<br>Tr. Start | Duration of<br>Antitumor<br>Treatment<br>(months) | Time since Previous Antitumor Treatment (months) | Setting | Туре |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXX | 1 | ddmmmyyyy | NA | XX.X | XXX.X | | Primary Tumor | Surgery |
| | | 2 | ddmmmyyyy | mmmyyyy | xx.x * | XXX.X * | XX.X * | Adjuvant | Chemotherapy |
| | | | | | | | | | Radiation Therapy |
| XXXX | XXXX | 1 | | | | | | | •••• |
| | | | | | | | | •••• | •••• |

Only patients with at least one therapy are displayed.

NA= Not Applicable

Weeks to Tr. Start: from antitumor treatment/procedure stop date to treatment start date.

Duration of Antitumor Treatment (weeks): from start date to stop date.

Time since previous Antitumor Treatment (weeks): from stop date of previous line (chron. seq.) to start date of current line.


[Program Path; Date/Time Produced; Date Data Extract]

### <u>Programming notes:</u>

Sort by pt no., chron. seq. number.

Select only patients with prior antitumor treatments/procedures = 'yes' or derived 'yes'.

<sup>\*:</sup> Estimated time when incomplete date was reported

Appendix 3.4.6 - Demography and Pretreatment: Tumor History - Prior Systemic Therapies - Treated Patients -

#### Page by Regimen

| Pt.<br>No. | Chron Seq.<br>No. | Setting | Drug<br>Name | Dose /<br>Unit /<br>Schedule | Start Date | Stop Date | Duration of<br>treatment<br>(months) | Best<br>Response | Response Date | Relapse / Progression<br>Date |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 2 | Primary Tumor | xxxxxxxx | | ddmmmyyyy | ddmmmyyyy | XXX.X | CR | ddmmmyyyy | ddmmmyyyy |
| | 3 | Metastatic | XXXXXXX | | ddmmmyyyy | ddmmmyyyy | XXX.X | | NA | NA |
| XXXX | 1 | Primary Tumor | XXXXXXX | XXXXXXX | ddmmmyyyy | mmyyyy | xxx.x* | PR | ddmmmyyyy | mmyyyy |
| | 2 | - | XXXXXXX | XXXXXXX | | | | | | |
| | n | | | | | | | | | |
| XXXX | 1 | | XXXXXXX | | ddmmmyyyy | ddmmmyyyy | XXX.X | | | |

Only patients with at least one therapy are displayed.

Best Response: CR= Complete Response, PR= Partial Response, SD= Stable Disease, PD = Progressive Disease, NE=Not Evaluable, NAS= Not Assessed, NA= Not Applicable.

\*: Estimated time when incomplete date was reported


[Program Path; Date/Time Produced; Date Data Extract]

### <u>Programming notes:</u>

Sort by pt no., chron. seq. number.

Select only patients with systemic therapy ='yes' or derived 'yes'.

Start/Stop Date: correspond to start/stop date in the header page when for the given Chron. Seq No. the variable Type can be linked to "Systemic Therapy" (see ALG document for derivation)

Appendix 3.4.7 – Demography and Pretreatment: Tumor History - Prior Surgeries - Treated Patients –

## Page by Regimen

| Pt. No. | Primary diagnosis | Chron.<br>Seq. No. | Setting | Date | Surgical<br>Procedure |
|---|---|---|---|---|---|
| XXXX | XXXX | 1 | Primary Tumor | ddmmmyyyy | xxxxxxxxxxxxxxxxxx |
| | | 2 | Locally Advanced | ddmmmyyyy | xxxxxxxxxxxxxxxxxx |
| XXXX | XXXX | | | | |
| ••• | | 1 | ••• | | |
| | | | •••• | | |

Only patients with at least one surgery are displayed.


[Program Path; Date/Time Produced; Date Data Extract]

### Programming notes:

Sort by pt no., chron. seq. number.

Select only patients with any prior surgery ='yes' or derived 'yes'.

Date: corresponds to start date in the header page when for the given Chron. Seq No. the variable Type can be linked to "Surgery" (see ALG document for derivation)

Appendix 3.4.8 – Demography and Pretreatment: Tumor History - Prior Radiotherapies - Treated Patients –

## Page by Regimen

| Pt.<br>No. | Primary<br>Diagnosis | Chron.<br>Seq.<br>No. | Setting | Irradiated<br>BM (%) | Start Date | Stop Date | Irradiation<br>Site | Best<br>Response | Date of Best<br>Response | Date of<br>Progression |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXX | 1 | Primary<br>Tumor | XX.X | ddmmmyyyy | ddmmmyyyy | xxxxxxx | CR | ddmmmyyyy | ddmmmyyyy |
| | | 2 | Adjuvant | | | | XXXXXXX | | NA | ddmmmyyyy |
| | | | | | | | XXXXXXX | PR | ddmmmyyyy | NA |
| XXXX | XXXX | 1 | •••• | XX.X | mmmyyyy | mmmyyyy | XXXXXXX | | | |
| XXXX | XXXX | | | XX.X | ddmmmyyyy | ddmmmyyyy | XXXXXXX | | | |

Only patients with at least one radiotherapy are displayed.

Best Response: CR = Complete Response, PR= Partial Response, SD = Stable Disease, PD = Progressive Disease, NE= Not Evaluable, NAS= Not Assessed, NA = Not Applicable


[Program Path; Date/Time Produced; Date Data Extract]

## <u>Programming notes</u>:

Sort by pt no., chron. seq. number.

Select only patients with Prior Radiotherapies = 'yes' or derived 'yes'.

Start/Stop Date: correspond to start/stop date in the header page when for the given Chron. Seq No. the variable Type can be linked to "Radiotherapy" (see ALG document for derivation)

Appendix 3.4.9 - Demography and Pretreatment: General Medical History and Physical Examination Findings - Treated Patients -

## Page by Regimen

| Pt. No. | Age/Sex/Race | Primary Diagnosis | Medical Conditions /<br>Physical Findings | Status |
|---|---|---|---|---|
| XXXX | 38/M/W | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx | Active |
| | | | xxxxxxxxxxxxxxxxxxxxxxxx | Controlled |
| | | | xxxxxxxxxxxxxxxxxxxxxxxx | Past |
| XXXX | xx/x/x | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx | Past |
| XXXX | xx/x/x | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Active |

Only patients with at least one finding are displayed.

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming notes:

Sort by pt. no, status (Active, Controlled and Past)

Select only patients with medical history/physical findings = 'yes' or derived 'yes'.

## Appendix 3 – Section 5 – Treatment Exposure

Appendix 3.5.1 – Treatment Exposure: Treatment Administration Details - Treated Patients -

### Page by Regimen

| Pt.<br>No. | Cycle | Tr.<br>Delay | Dose<br>Reduced<br>at Cycle<br>Start | Intra Cycle<br>Modification | Dose<br>Level<br>(mg/day) | BSA<br>(m2) | Day | Taken Dose (mg) | Date of Admin. | Time of Admin. |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | Cy 1 | | | Y | XXX.X | X.XX | 1 | XXX.X | ddmmmyyyy | hh:mm |
| | | | | | | | | XXX.X | | hh:mm |
| | | | | | | | 5 | | ddmmmyyyy | |
| | | | | | | | •••• | | | |
| | | | | | | | 7 | | | |
| | Cy 2 | Y | Y | | XXX.X | X.XX | 1 | XXX.X | ddmmmyyyy | hh:mm |
| | | | | | | | | ••• | ••• | ••• |
| XXX | Cy 1 | | | | | X.XX | 1 | XXX.X | ddmmmyyyy | hh:mm |

[Protocol No.; Study Description] [Program Path; Date/Time Produced; Date Data Extract]

### **Programming Notes:**

Sort by pt. no., study period, day, date of administration.

## Appendix 3.5.2 – Treatment Exposure: Reasons for Treatment Delay, Dose Reduction - Treated Patients -

### Page by Regimen

| Pt<br>No. | Cycle | Cycle<br>Duration<br>(weeks) | Trt.<br>Delay | Reason | Specify | Dose<br>Reduced at<br>cycle start | Reason | Specify | Intra-cycle<br>Modification | Reason | Specify | Dose<br>Level<br>(mg/day) | Day | Taken<br>Dose<br>(mg) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | Cy 1 | XX.XX | | | | | | | | xxxxxxxx | | XXX.X | 1 | XXX.X |
| | | | | | | | | | | | | | ••• | XXX.X |
| | | | | | | | | | | | | | 5 | XXX.X |
| | Cy 2 | XX.XX | | | | Y | (H) | xxxxxx | | xxxxxxxx | | XXX.X | 1 | xxx.x |
| | | •••• | | | | | | | | | | | | ••• |
| | Cy n | xx.xx<br>(xx.xx) | | | | | | | | | | | | ••• |
| xxxx | Cy 1 | XX.XX | Yes | (N-H) | xxxxxx | | | | Yes | | | ••• | 1 | XXX.X |
| | | ••• | | | | ••• | | | | | | | ••• | •••• |

Only patients/cycles for whom any treatment modifications are reported.

Duration of the last cycle of treatment is calculated from last cycle start date to end of treatment date; the per-protocol cycle duration is reported within brackets Reason for Intra Cycle Modification includes Reason for Dose Omitted and Dose Reduced Intra Cycle.

Reasons: H=Hematological toxicity, N-H=Non-Hematological toxicity, O=Other, specify.


[Program Path; Date/Time Produced; Date Data Extract]

### **Programming Notes:**

Sort by pt. no., study period, day. Select only patients for whom any modification applies, i.e. either treatment delay=Y or Dose reduced at cycle start=Y or intra-cycle modification=Y.

Appendix 3.5.3 – Treatment Exposure: Dose Intensity and Cumulative Dose
- Treated Patients –

Page by Regimen

Intended Dose Intensity (mg/wk): xxx.x

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study Period | No. of<br>Days of<br>Treatment | Taken Dose (mg) | BSA<br>(m2) | %<br>Scheduled<br>Dose | Treatment<br>Duration<br>(weeks) | Absolute<br>D.I.<br>(mg/wk) | Relative<br>D.I.<br>(%) | Progressive<br>Cum. Dose<br>(mg) |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | 38/F/W | Cy 1 | XX | XXX.X | X.XX | XX.X | XX.X | XXX.X | XX.X | XXX.X |
| | | Cy 2 | XX | XXX.X | | XX.X | XX.X | XXX.X | XX.X | XXX.X |
| | | Cy x | XX | XXX.X | X.XX | XX.X | xx.x(3) | XXX.X | XX.X | XXX.X |
| | | Whole Period | | | | | XX.X | XXX.X | XX.X | XXX.X |
| XXXX | xx/x/x | Cy 1 | XX | XXX.X | X.XX | XX.X | XX.X | XXX.X | XX.X | XXX.X |
| | | Cy 2 | XX | XXX.X | | XX.X | XX.X | XXX.X | XX.X | XXX.X |
| | | Cy x | XX | XXX.X | X.XX | XX.X | xx.x(3) | XXX.X | XX.X | XXX.X |
| | | Whole Period | | | | | XX.X | XXX.X | XX.X | XXX.X |

Race: W= White, B= Black, A= Asian, O= Not listed, N= Not allowed to ask per local regulation.

% Scheduled Dose: the ratio between dose (mg) and intended dose x 100.

Treatment Duration for last cycle and whole period: from the last cycle start date or from first dose date respectively, to end of treatment date. Duration reported in brackets is used for dose intensity calculation and considers the per protocol cycle duration.

Relative D.I.: the ratio between absolute dose intensity and intended dose intensity x 100.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by pt. no., study period.

## Appendix 3.5.4 – Treatment Exposure: Pharmacokinetics Blood Sampling Time - Treated Patients –

## Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Tr.<br>Admin<br>Date | Tr.<br>Admin.<br>Time | Study Day | Study<br>Time | Specimen<br>Collection<br>Date | Specimen<br>Collection<br>Time |
|---|---|---|---|---|---|---|---|---|
| XXXX | 52/F/W | Cy 1 | ddmmmyyyy | hh:mm | 1 | 1 | ddmmmyyyy | hh:mm |
| | | | | | | 2 | ddmmmyyyy | hh:mm |
| | | | | | | 3 | ddmmmyyyy | hh:mm |
| | | | ddmmmyyyy | hh:mm | X | ••• | ••• | ••• |
| xxxx | xx/x/x | Cy 1 | ddmmmyyyy | hh:mm | 1 | | ddmmmyyyy | hh:mm |
| | | | • • • | | | | • • • | |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by pt. no., study period, tr. Admin. date, study day, study time, collection date, collection time.

Study day is the one indicated on the PK form of the CRF.

## Appendix 3 – Section 6 – Treatment Efficacy

Appendix 3.6.1 - Treatment Efficacy - Target and Non Target Lesions by Assessment Visit - Treated Patients -

Page by Regimen

| Pt.<br>No. | Study<br>Period | Date | Days<br>to/from<br>Tr. Start | Les.<br>Type | Les.<br>No. | Lesion<br>Description | Eval.<br>(Y/N) | Lymph<br>Node | Prior<br>Loco-<br>regionally<br>Treated<br>Lesion | New<br>Les. | N.<br>A. | Method | Target L.<br>Measure<br>(mm) | Target L. % Change from Pretr | Target<br>L.<br>Nadir | Target.L.<br>% Change<br>from Nadir | Non<br>Target<br>L.<br>Status |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Pretr. | ddmmmyyyy | XXX | T | XX | XXXXXXXXX | | Y | Y | | | XX | XXXX | | | | |
| | | | | | XX | XXXXXXX | | | | | | XX | XXXX | | | | |
| | | | | | | All Target L. | | | | | | | XXXX | | | | |
| | | | | NT | XX | XXXXX | | | | | | ••• | | | | | |
| | Onc 1 | ddmmmyyyy | XXX | T | XX | XXXXXXXXX | Y | Y | | | | XX | XXXX | | | | |
| | | | | | XX | XXXXXXX | Y | | | | | XX | XXXX | $\pm xxx.x$ | | | |
| | | | | | XX | XXXXXXX | Y | | | Y | | XX | XXXX | | | | |
| | | | | | | All Target L | Y | | | | | | XXXX | $\pm xxx.x$ | Y | | |
| | | ddmmmyyyy | XXX | NT | XX | XXXXXXX | | | | | | | | | | | Α |
| | Onc x | ddmmmyyyy | XXX | T | | ••• | | | | | | | | | | | |
| | | | | | | All Target L | Y | | | | | | XXXX | $\pm xxx.x$ | | XXXX | |
| XXX | Pretr. | ddmmmyyyy | XXX | T | XX | XXXXXXXXX | | | | | | XX | XXXX | | | | |
| | | | | | | All Target L. | | | | | | | XXXXX | | | | |
| | Onc. 1 | ddmmmyyyy | XXX | T | XX | XXXXXXXXX | N | | | | | xx* | XXXX | | | | |
| | | | | | | All Target L | N | | | | | | XXXX | | | | |

Lesion Type: T=Target Lesion, NT=Non Target Lesion

Eval (Y/N): a target lesion is not considered as evaluable if missing measure and/or method, or method different from pretreatment assessment; the set of all target lesions is not evaluable if even one only target lesion is not evaluable.

N.A.: Not Assessed.

Method: 1=Physical Exam. (measurement by caliper), 2=X-ray, 3=Echo/Ultrasounds, 4=CT scan, 5=Scintigraphy, 6=MRI/NMR, 7=Linear Tomography, 8=Photography, 10=Bronchoscopy, 13=Spiral CT-Scan, 14=PET, 15=MIBG Scan, 16=99tc Scan, 17=MR Spectroscopy, 18=Thallium Spectroscopy, 19=Angiography, 20=Bone Scan, 98=Other, specify in the Physician's Comments page. Methods different from the pretreatment one are marked by '\*'.

Non Target Lesions: Status: A=Absent (CR); P=Present (Non-CR/Non-PD); UPD=Unequivocal Progressive Disease.

Nadir: lowest value of All Target Lesions throughout the whole study period, baseline included. %Change from Nadir: only for study periods following the period when the nadir is reported.


[Program Path; Date/Time Produced; Date Data Extract]

<u>Programming Notes:</u> Sort by pt. no., study period, les type (T, NT), les. no..

## Appendix 3.6.2 - Treatment Efficacy - Response Status by Assessment Visit - Treated Patients -

#### Page by Regimen

| | | | | | | | | If CR | or PR |
|---|---|---|---|---|---|---|---|---|---|
| Pt.<br>No. | Study<br>Period | Assessment<br>Date | Days<br>from<br>Tr.<br>Start | Response | Response<br>Status | Date of<br>Documented<br>PD | Weeks to<br>PD | First Response<br>Date | Response<br>Confirmation<br>Date |
| XXX | One 1 | ddmmmyyyy | XXX | Target Lesion | CR | | | | _ |
| | | | | Non Target Lesion | NE | | | | |
| | | | | Overall | PR | | | | |
| | One 1 | ddmmmyyyy | XXX | ••• | | ••• | ••• | ••• | ••• |
| | | | | Overall | PD | ddmmmyyyy | XXX.X | | |
| | Best OR | | | Best Overall | PR | | | ddmmmyyyy | ddmmmyyyy* |
| XXX | One 1 | | | | XX | | | | |
| | ••• | ••• | | | ••• | | | | |
| | One 3 | | | | XX | ddmmmyyyy | XXX.X | | |
| | Best OR | | | Best Overall | CR | ••• | | ddmmmyyyy * | ddmmmyyyy |

Assessment date: the date of the first tumor lesion assessment in the relevant study period.

Response Status: CR = Complete Response, PR = Partial Response, SD = Stable Disease, NCR/NPD= Non-CR/Non-PD, UPD= Unequivocal PD, PD = Progressive Disease, NE= Not Evaluable, NA = Not Applicable.

Date of Documented PD was derived as the first tumor lesion assessment date in the relevant study period. Weeks to PD: from the first treatment date to the date of documented PD. First Response Date: when not recorded on CRF, the \* indicates that the date was derived as the latest date among all tumor lesion assessment dates at the first visit when a response (CR or PR) was reported. Response Confirmation Date: when not recorded on CRF, the \* indicates that the date was derived as the latest date among all tumor lesion assessment dates at the second visit when a response (CR or PR) was reported.


[Program Path; Date/Time Produced; Date Data Extract]

<u>Programming Notes:</u> Sort by pt. no., study period, les type (target, non-target, overall).

Appendix 3.6.3 - Treatment Efficacy – Best Overall Response and Time to Progression, Progression Free Survival, Overall Survival, Response Duration and Stable Disease Duration
- Treated Patients -

Page by Regimen/Assigned Dose Level (mg/m2/day): <xi >

| Pt.<br>No | Pt.<br>Evaluable<br>for<br>Efficacy<br>(Y/N) | Tr. Start<br>Date | Total<br>No. of<br>Cycles | Dose<br>Intensity<br>(mg/wk) | | Date of<br>First<br>Response | Date of PD | Date of<br>Death | Last Onc.<br>Assessment<br>Date | Last<br>Recorded<br>Date | TTP (days) | OS<br>(days) | PFS (days) | Response<br>Duration<br>(days) | Stable<br>Disease<br>Duration<br>(days) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Y | ddmmmyyyy | 4 | XXX.X | CR | ddmmmyy | | ddmmmyyyy | ddmmmyyyy | | xxx.x + | | XXX.X | xxx.x + | |
| XXX | Y | ddmmmyyyy | 3 | XXX.X | SD | | ddmmmyyyy | | ddmmmyyyy | ddmmmyyyy | XXX.X | xxx.x + | XXX.X | | XXX.X |
| XXX | Y | ddmmmyyyy | X | XXX.X | PR | ddmmmyy<br>* | 7 | | ddmmmyyyy | ddmmmyyyy | xxx.x + | xxx.x + | xxx.x + | xxx.x + | |
| XXX | Y | ddmmmyyyy | X | XXX.X | PD | | ddmmmyyyy | | ddmmmyyyy | ddmmmyyyy | XXX.X | xxx.x + | XXX.X | | |
| XXX | N | ddmmmyyyy | X | XXX.X | CR | ddmmmyy | | | ddmmmyyyy | ddmmmyyyy | xxx.x + | xxx.x + | xxx.x + | xxx.x + | |
| XXX | | ddmmmyyyy | X | XXX.X | SD | | | ddmmmyyyy | ddmmmyyyy | | XXX.X | | XXX.X | | XXX.X |
| XXX | Y | ddmmmyyyy | X | XXX.X | SD | | | ddmmmyyyy | ddmmmyyyy | | xxx.x + | | XXX.X | | xxx.x + |

Best Overall Response: as reported by the investigator at the completion of treatment; CR = Complete Response, PR = Partial Response, SD = Stable Disease, PD = Progressive Disease, NE= Not Evaluable.

Date of First Response: when not recorded on CRF, the \* indicates that the date was derived as the latest date among all tumor lesion assessment dates at the first visit when a response (CR or PR) was reported.

Last Recorded Date: for patients still alive it is the last available date in CRF.

(+): indicates censored time.


[Program Path; Date/Time Produced; Date Data Extract]

### <u>Programming Notes</u>:

Sort by pt. no.

D.I.: the dose intensity to be reported is the one calculated for the whole treatment period.

# Appendix 3.6.4 – Treatment Efficacy: ECOG Performance Status - Treated Patients -

Page by Regimen

| Pt.<br>No. | Study<br>Period | Date | Study<br>Day | ECOG<br>PS |
|------------|-----------------|-----------|--------------|------------|
| XXXXXX | Pretr. | ddmmmyyyy | | 3 § |
| | Cy 1 | ddmmmyyyy | 1 | 0 |
| | ••• | • • • • | •••• | •••• |
| | Cy n | ddmmmyyyy | 1 | |

At pretreatment: Performance Status >1 is identified by § (violation of inclusion criterion 05).


[Program Path; Date/Time Produced; Date Data Extract]

Programming Notes:

Sort by pt. no., study period, date.

## *Appendix 3 – Section 7 – Adverse Events*

Appendix 3.7.1 – Adverse Events: All Reported Adverse Events by Assessment Visit and AE MedDRA Preferred Term
- Treated Patients -

### Page by Regimen

| Pt.<br>No. | Study<br>Period | Cycle Start<br>Date | Adverse<br>Event | CTC<br>Grade | Serious | Start Date | A.<br>P. | Stop Date | S.<br>P. | Rel.<br>to<br>Study<br>Proc. | Rel.<br>to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease | Action<br>Taken | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | Pretr. | | XXXXXXXXX | 1 | N | ddmmmyyyy | | ddmmmyyyy | | Y | | N | | R |
| | | | XXXXXXXXX | 1 | N | | Y | | Y | N | | N | | NR |
| | | | XXXXXXXXX | 2 | | | Y | ddmmmyyyy | | N | | Y | | R |
| | Cy 1 | ddmmmyyyy | XXXXXXXXX | X | | | Y | | Y | | No | | No | NR |
| | | | XXXXXXXXX | | | ddmmmyyyy | | | Y | | Un | N | No | NR |
| | | | xxxxxxxxx | 3 | Y | ddmmmyyyy | | ddmmmyyyy | | | Po | Y | D/C | R |
| | ••• | ••• | • • • | | | ••• | | ••• | | | | ••• | | ••• |

AP/SP: Already present/Still present.

Related to Study Treatment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.

Action Taken: No=None; D/C=Dose Delayed/Changed; PW=Drug Permanently Withdrawn.

Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.

[Protocol No. (Study Description)]

[Program Path; Date/Time Produced; Date Data Extract]

### Programming Notes:

Sort by pt. no., study period, AE MedDRA Preferred Term, AE page no., AE seq no.. Include also records of End of Adverse Events Reporting Period and of Follow-up.

Appendix 3.7.2 - Adverse Events: Adverse Events Related to Study Procedure at Pretreatment - Treated Patients -

## Page by Regimen

| Pt. No. | Adverse Event | CTC<br>Grade | Serious | Start Date | A.<br>P. | Stop Date | S.<br>P. | Rel. to Study<br>Procedure | Rel. to Study<br>Disease | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXXXX | X | N | ddmmmyyyy | | ddmmmyyyy | | Y | N | |
| | XXXX | X | N | | | | | | N | |
| | xxxxxxx xxxx xxx | X | N | | Y | | | | Y | R |
| | XXXXXXX | X | N | ddmmmyyyy | | | Y | | ••• | NR |
| XXXX | ••• | | | ••• | | ••• | | | N | |
| | | | ••• | | | ••• | | | Y | |

Only AEs reported at pretreatment visit and related to study procedure are displayed.

AP/SP: Already present/Still present.

Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.


[program path; date/time produced; date data extract]

#### Programming Notes:

Sort by pt. no., study period, AE MedDRA Preferred Term, AE page no., AE seq. no.

Select only records at pretreatment and with variable "Related to study procedure" =Y or missing

## Appendix 3.7.3 – Adverse Events: Serious Adverse Events - Treated Patients -

### Page by Regimen

| Pt.<br>No. | Adverse<br>Event | Study<br>Period | Cycle<br>Start Date | Serious | CTC<br>Grade | Start Date | A.<br>P. | Stop Date | S.<br>P. | Rel. to<br>Study<br>Proc. | Rel. to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease | Action<br>Taken | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXXXXXXX | Pretr. | | | 2 | ddmmmyyyy | | ddmmmyyyy | | N | | N | | R |
| | | Cy 1 | ddmmmyyyy | | 3 | ddmmmyyyy | | | | | De | Y | D/C | NR |
| | | | | Y | 4 | | Y | | Y | | Pr | Y | D/C | R |
| | | Cy x | ddmmmyyyy | Y | | ••• | Y | ddmmmyyyy | | | | ••• | PW | |
| | xxxxxxxxx | Cy 1 | ddmmmyyyy | | 1 | ddmmmyyyy | | ddmmmyyyy | | | | Y | No | NR |
| | | | | | | ddmmmyyyy | | | Y | | Po | | | R |
| | | Cy x | ddmmmyyyy | Y | | | Y | ddmmmyyyy | | | | | | NR |
| XXXX | ••• | | | | | ••• | | ••• | | | | | | |

All occurrences of AEs that were reported as Serious at least once for the patient in the course of the study are displayed.

AP/SP: Already present/Still present.

Related to Study Treatment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.

Action Taken: No=None; D/C=Dose Delayed/Changed; PW=Drug Permanently Withdrawn.

Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by pt. no., AE MedDRA Preferred Term, study period, AE page no., AE seq no..

Select AE Preferred terms that had the variable 'Serious'=Y at least once within the patient in the course of the study, including pretreatment, End of Adverse Events Reporting Period and of Follow-up.

## Appendix 3.7.4 – Adverse Events: Adverse Events with CTC Grade 3 to 5

#### Page by Regimen

| Pt.<br>No | Adverse<br>Event | Study<br>Period | Cycle Start<br>Date | CTC<br>Grade | Serious | Start Date | A.<br>P. | Stop Date | S.<br>P. | Rel. to<br>Study<br>Proc | Rel. to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease | Action<br>Taken | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | XXXXXXXX<br>XX | Pretr. | | 3 | N | ddmmmyyyy | | ddmmmyyyy | | | No | Y | No | R |
| | XXXXXXX<br>XX | Cy 1 | ddmmmyyyy | 3 | N | | Y | | Y | | Un | Y | D/C | NR |
| | | <br>Cy x | ddmmmyyyy | | Y<br> | | <br>Y | | <br>Y | | Pr<br>Pr | N<br>N | <br>No | <br>NR |
| | XXXXXXXX<br>XX | Cy 1 | ddmmmyyyy | ••• | | ddmmmyyyy | | | Y | | Un | Y | No | NR |
| | | <br>Cy x | ddmmmyyyy | 4 | Y | ddmmmyyyy | | ddmmmyyyy | | | De | Y | D/C | R<br> |

Only AE occurrences at the time when CTC grade > 2 are displayed.

AP/SP: Already present/Still present.

Related to Study Treatment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.

Action Taken: No=None; D/C=Dose Delayed/Changed; PW=Drug Permanently Withdrawn.

Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.


[Program Path; Date/Time Produced; Date Data Extract

#### **Programming Notes:**

Sort by pt. no., study period, AE MedDRA Preferred Term, AE page no., AE seq. no..

Selct only the occurrences of AEs when CTC grade > 2. Include also occurrences reported with grade > 2 at pretreatment or at End of Adverse Events Reporting Period or at Follow-up.

Appendix 3.7.5 – Adverse Events: Patients with Adverse Events Leading to Withdrawal from Study Treatment - Treated Patients -

### Page by Regimen

| Pt.<br>No. | Adverse<br>Event | Study<br>Period | Cycle<br>Start Date | CTC<br>Grade | Serious | Start Date | A.<br>P. | Stop Date | S.<br>P. | Rel. to<br>Study<br>Proc. | Rel. to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease | Action taken | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXXXXXXX | Pretr. | | 2 | | ddmmmyyyy | | ddmmmyyyy | | N | | N | | R |
| | | Cy 1 | ddmmmyyyy | 3 | Y | ddmmmyyyy | | | | | De | Y | D/C | NR |
| | | | | 4 | Y | | Y | | Y | | Pr | Y | D/C | R |
| | | Cy x | ddmmmyyyy | | N | ••• | Y | ddmmmyyyy | | | | | PW | ••• |
| | XXXXXXXXX | Cy 1 | ddmmmyyyy | 1 | | ddmmmyyyy | | ddmmmyyyy | | | | Y | No | NR |
| | | | | | | ddmmmyyyy | | | Y | | Po | | | R |
| | | Cy x | ddmmmyyyy | ••• | ••• | | Y | ddmmmyyyy | | | ••• | ••• | | NR |
| XXXX | | | | | | ••• | | | | | | | | |

Only patients that had at least one AE whose Action Taken was Drug Permanently Withdrawn are displayed.

AP/SP: Already present/Still present.

Related to Study Treatment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.

Action Taken: No=None; D/C=Dose Delayed/Changed; PW=Drug Permanently Withdrawn.

Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Sort by, pt. no., study period, AE MedDRA Preferred Term, AE page no., AE seq no..

Select patients that had at least one AE whose Action Taken was Drug Permanently Withdrawn. Of these patients report all AEs.

Include also records of End of Adverse Events Reporting Period and of Follow-up.

## Appendix 3.7.6 – Adverse Events: End of AE Reporting Period and Follow-Up - Treated Patients –

## Page by Regimen

| Pt.<br>No | Tr. Last<br>Date | Study<br>Period | Adverse<br>Event | CTC<br>Grade | Serious | Start Date | A.<br>P. | Stop<br>Date | S.<br>P. | Rel. to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease | Outcome | If Ongoing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | ddmmmyyyy | AE End | XXXXXXXXX | X | N | | Y | | Y | No | N | NR | Chronic/Stable |
| | | | XXXXXXX | X | N | | Y | | Y | Un | Y | NR | Continue to follow |
| | | | xxxxxxxxx | X | | ddmmmyyyy | | | Y | Po | N | NR | New Anticancer therapy |
| xxxx | ddmmmyyyy | AE FU1 | § xxxxxxx | X | | | Y | | Y | De | N | NR | Chronic/Stable |

• •

AEs not recovered in Follow-up are identified by §.

AP/SP: Already present/Still present.

Related to Study Treatment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite. Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.


[Program Path; Date/Time Produced; Date Data Extract

#### **Programming Notes:**

Sort by pt. no., study period, AE MedDRA Preferred Term, AE page no., AE seq. no..

Select AEs with study period = 'End of AE reporting period' or 'Follow-up'.

Appendix 3.7.7 – Adverse Events: All Reported Adverse Events by System Organ Class, AE MedDRA Preferred Term and Investigator's Term - Treated Patients -

## Page by Regimen

| Pt. No. | System<br>Organ Class | Adverse Event | Investigator's Term | Study Period | Cycle<br>Start Date | CTC<br>Grade | Serious | Rel. to<br>Study<br>Proc. | Rel. to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXXXXXXXXX | XXXXXXXXXXXX | XXXXXXXXXXXX | Pretr. | | X | N | N | De | |
| | | XXXXXXXXXXX | XXXXXXXXXXXX | Cy 1 | ddmmmyyyy | X | Y | | Pr | Y |
| | | XXXXXXXXXXXX | XXXXXXXXXXXX | Су х | ddmmmyyyy | X | N | | • • • | ••• |
| | | | XXXXXXXXXXXX | Су х | ddmmmyyyy | X | N | | | Y |
| | | | | Cy 1 | ddmmmyyyy | X | ••• | | Po | |
| | | | | Су х | ddmmmyyyy | X | ••• | | | |
| XXXXX | XXXXXXXXXXX | XXXXXXXXXXXX | XXXXXXXXXXXX | ••• | | X | | | | |
| | | XXXXXXXXXXXX | XXXXXXXXXXXX | ••• | | X | | | | |

Related to Study Treatment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Sort by pt. no., System Organ Class, AE MedDRA Preferred Term, AE Investigator's Term, study period, AE page no., AE seq no..

## Appendix 3.7.8 – Adverse Events: Hospitalization - Treated Patients -

## Page by Regimen

| Pt.<br>No. | Age/Race<br>/Sex | Tr. Start<br>Date | Tr. Last<br>Date | Reason | Description | Date of<br>Admission | Date of<br>Discharge | Ongoing | Duration (days) | Weeks<br>from<br>Tr. Start |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | 35/W/M | ddmmmyyyy | ddmmmyyyy | Adverse | | ddmmmyyyy | ddmmmyyyy | | XXX | XXX |
| | | 5555 | 5555 | event | | | | | | |
| | | | | Progressive | | ddmmmyyyy | | V | | XXX |
| | | | | Disease | | ddiiiiiiiyyyy | | 1 | | |
| xxxx | xx/x/x | ddmmmyyyy | ddmmmyyyy | Instrumental procedure | | ddmmmyyyy | | Y | | XXX |
| XXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | Other | XXXXXXXXXXXX | ddmmmyyyy | ddmmmyyyy | | XXX | XXX |

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.

Duration (days): from date of admission to date of discharge.

Weeks from Tr. Start: from treatment start date to date of admission.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by pt. no., admission date, seq. no.

Appendix 3.7.9 – Deaths - Treated Patients -

## Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Tr. Start<br>Date | Tr. Last<br>Date | Total<br>No. of<br>Cycles | Cumulative<br>Dose<br>(mg/m2) | Date of<br>Death | CRF<br>Source | Days<br>from Tr.<br>Last Date | Most<br>Probable<br>Cause | Details | Investigator<br>Causality<br>Assessment |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 38/M/W | ddmmmyyyy | ddmmmyyyy | 2 | XXXX.X | ddmmmyyyy | FU | XXX | PD | | Un |
| XXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | X | XXXX.X | ddmmmyyyy | Death | xxx* | AΕ | XXXXXXXXX | No |
| XXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | X | XXXX.X | ddmmmyyyy | Death | XXX | Other | XXXXXXXXX | Po |
| XXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | X | XXXX.X | ddmmmyyyy | AΕ | XXX | AΕ | XXXXXXXX | Pr |
| XXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | X | XXXX.X | ddmmmyyyy | AΕ | XXX | ΑE | | ••• |
| XXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | X | XXXX.X | ddmmmyyyy | ΑE | XXX | | | |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

CRF Source: (Death): Death date reported in Death Form, (FU): Death date reported in Survival Follow-up Form, (AE): Death date reported in AE Form.

Days from treatment last date: \* if <= 28 days.

Investigator Causality Assessment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by pt. no..

## Appendix 3.7.10 – Deaths: Autopsy Result - Treated Patients –

## Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Days from Tr. Last Date to Death Date | Most Probable Cause | Details | Investigator<br>Causality<br>Assessment | Autopsy<br>Performed | Autopsy<br>Date | Autopsy<br>Result |
|---|---|---|---|---|---|---|---|---|
| xxxx | 38/M/W | XXX | Progressive Disease | | Pr | Y | ddmmmyyyy | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| xxxx | xx/x/x | xxx* | Adverse Event | | Po | Y | ddmmmyyyy | |
| XXXX | xx/x/x | XXX | Other | xxxxxxxxxx | | N | | |
| XXXX | xx/x/x | XXX | | | | N | | |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

Days from treatment last date to death date: \* if <= 28 days.

Investigator Causality Assessment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by pt. no..

### Appendix 3 - Section 8 – Laboratory Assessments

Appendix 3.8.1 – Laboratory Assessments: Hematology by Laboratory Test, Patient and Study Period - Treated Patients -

Page by Regimen /Laboratory Test: < e.g. Neutrophils >

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Cycle<br>Start Date | Date of Sampling | Study<br>Day | Collected<br>Value | Collected<br>Unit | L/H | Converted<br>Value | Converted<br>Unit | CTC<br>Grade |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 52/F/W | Pretr. | | ddmmmyyyy | -XX | XXX.XX | XXXX | L | XXX.XX | XXXX | X |
| | | Cy x | ddmmmyyyy | ddmmmyyyy | XX | ••• | | | ••• | | 3 * |
| | | | | | XX | | ••• | ••• | ••• | | 4 * |
| | | ••• | | ••• | ••• | ••• | | • • • | ••• | | |
| XXXX | | Pretr. | | ddmmmyyyy | XX | | | • • • | | | 2 |
| | | | ••• | ••• | | ••• | | | ••• | • • • | |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

Converted Unit: either the unit reported in the NCI CTCAE v3.0 or the Conventional Unit, depending on the analyzed lab test.

CTC Grade - NCI CTCAE v3.0: N= Not Applicable, U= Unknown. The '\*' identifies the occurrence(s) of CTC grades= 3 or 4.

L/H: Below/Above Normal Limits.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Sort by "page by variables", pt. no, study period, date of sampling, study day. If feasible lab test is to be ordered as per CRF appearance.

The listing must include all the hematological labs (including also the ones that are not listed in the NCI CTCAE v.3.0).

Appendix 3.8.2 – Laboratory Assessments: Blood Chemistry by Laboratory Test, Patient and Study Period
- Treated Patients -

Page by Regimen /Laboratory Test: < e.g. ALT >

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Cycle Start<br>Date | Date of Sampling | Study<br>Day | Collected<br>Value | Collected<br>Unit | Collected<br>Lower<br>Limit | Collected<br>Upper<br>Limit | L/H | Converted Value | Converted<br>Unit | CTC<br>Grade |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 52/F/W | Pretr. | | ddmmmyyyy | - XX | XXX.XX | XXX.XX | XXX.XX | XXX | L | XXX.XX | XXXX | N |
| | | | | | | XXX.XX | XXX.XX | XXX.XX | XXX | | | | N |
| | | Cy x | ddmmmyyyy | ddmmmyyyy | XX | XXX.XX | XXX.XX | XXX.XX | XXX | Н | | | 3* |
| | | | | | | ••• | ••• | ••• | ••• | • • • | ••• | ••• | |
| | | | | ddmmmyyyy | XX | ••• | | | | L | | | 4* |
| | | | | ••• | | ••• | ••• | ••• | | | | | |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

Converted Unit: either the unit reported in the NCI CTCAE v3.0 or the Conventional Unit, depending on the analyzed lab test.

CTC Grade - NCI CTCAE v3.0: N= Not Applicable, U= Unknown. The '\*' identifies the occurrence(s) of CTC grades= 3 or 4.

L/H: Below/Above Normal Limits.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by "page by variables", pt. no, study period, date of sampling, study day.

If feasible lab test is to be ordered as per CRF appearance.

The listing must include all the biochemistry labs (including also the ones that are not listed in the NCI CTCAE v.3.0).

Appendix 3.8.3 – Laboratory Assessments: Coagulation by Patient, Study Period and Laboratory Test - Treated Patients –

### Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Cycle Start<br>Date | Date of Sampling | Study<br>Day | Laboratory<br>Test | Collected<br>Value | Collected<br>Unit | Collected<br>Lower<br>Limit | Collected<br>Upper<br>Limit | L/H | Converted<br>Value | Converted<br>Unit | CTC<br>Grade |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 52/F/W | Pretr. | | ddmmmyyyy | - xx | aPTT | XXX.XX | XXX.XX | XXX.XX | XXX | L | XXX.XX | XXXX | 2 |
| | | | | | | INR | XXX.XX | XXX.XX | XXX.XX | XXX | | ••• | | 1 |
| | | | | ddmmmyyyy | | aPTT | XXX.XX | XXX.XX | XXX.XX | XXX | Н | | | 2 |
| | | | | | | INR | XXX.XX | XXX.XX | XXX.XX | XXX | Н | ••• | ••• | 2 |
| | | Cy x | ddmmmyyyy | ddmmmyyyy | XX | ••• | ••• | ••• | ••• | ••• | | ••• | ••• | |
| | | | | 1.1 | | ••• | ••• | ••• | ••• | ••• | • • • | ••• | ••• | |
| | | | | ddmmmyyyy | XX | ••• | | ••• | ••• | | • • • • | | | |
| | | | | | | ••• | ••• | ••• | ••• | ••• | • • • | | | |
| | | | | ••• | | ••• | | ••• | ••• | | • • • | | | |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

Converted Unit: either the unit reported in the NCI CTCAE v3.0 or the Conventional Unit, depending on the analyzed lab test.

CTC Grade - NCI CTCAE v3.0: N= Not Applicable, U= Unknown. The '\*' identifies the occurrence(s) of CTC grades= 3 or 4.

L/H: Below/Above Normal Limits.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by pt. no, study period, date of sampling, study day, lab test.

If feasible lab test is to be ordered as per CRF appearance.

The listing must include all the coagulation labs (including also the ones that are not listed in the NCI CTCAE v.3.0).

## Appendix 3.8.4 – Laboratory Assessments: Urinalysis - Treated Patients –

## Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Cycle Start<br>Date | Date of Sampling | Study<br>Day | Laboratory<br>Test | Collected<br>Value |
|---|---|---|---|---|---|---|---|
| xxxx | 52/F/W | Pretr. | 44 | ddmmmyyyy | - XX | ph<br>glucose<br> | xx<br>negative<br>trace |
| | | Cy. 1 | ddmmmyyyy | ddmmmyyyy | XX | ph<br><br>protein | 1+ |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Sort by pt. no, study period, date of sampling, study day, lab test.

If feasible lab test is to be ordered as per CRF appearance.

Appendix 3.8.5 – Laboratory Assessments: Laboratory Normal Ranges of Hematological Tests

| Laboratory Test Description | Laboratory Test<br>Code | Sex | Age Min<br>(years) | Age Max<br>(years) | Lower Limit | Upper Limit | Unit |
|---|---|---|---|---|---|---|---|
| XXXXX | | Both | | | XXX.XX | XXX.XX | XXXXX |
| XXXXX | | | | | | ••• | |
| XXXXX | | Male | | | ••• | ••• | |
| XXXXX | | Both | | | ••• | ••• | |
| | | Female | | | | | ••• |
| ••• | | ••• | | | ••• | ••• | • • • |
| ••• | | ••• | | | ••• | ••• | • • • |
| ••• | | | | | ••• | ••• | • • • |

Normal ranges are not collected for hematological tests, Standard Normal Ranges expressed in Conventional Unit are used. Age class: age range 0-150 is a conventional range when lab. test normal ranges are valid for all ages


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by lab. Test (description, code), sex.

For each test belonging to WBC, report the unit expressed both in percentage and absolute count.

Appendix 3.8.6 – Laboratory Assessments: Laboratory Normal Ranges of Non-Hematological Tests - Treated Patients -

Page by: Laboratory Code: <xxxxx> Laboratory Name: <xxxxxxxxxxx>.

| Laboratory<br>Class | Assay | Initial Set (Y/N) | Date of Change | ate of Change Sex | | Age Max (years) | Lower Limit | Upper Limit | Unit |
|---|---|---|---|---|---|---|---|---|---|
| Blood | XXXXX | Y | | Male | XX | XX | XXX.XX | XXX.XX | |
| Chemistry | | | | | | | | | |
| | | | | | ••• | ••• | ••• | ••• | • • • |
| | | | | Female | XX | XX | | ••• | • • • • |
| | | | | | ••• | ••• | ••• | ••• | |
| XXXXXXXXXXX | XXXXX | N | ddmmmyyyy | Both | XX | XX | ••• | ••• | • • • |
| | | | | | ••• | ••• | ••• | ••• | |
| | XXXXX | | | | | | | ••• | |
| | | ••• | | | ••• | ••• | • • • | | |

Units are not converted, they are listed according to CRF reported units.

Age class: age range 0-150 is a conventional range when lab. test normal ranges are valid for all ages.


[Program Path; Date/Time Produced; Date Data Extract]

## **Programming Notes:**

Sort by "page by variables", laboratory class, assay, date of change, sex, age min.

Lab test ranges are not to be converted; they are to be listed according to the units reported on CRF.

## Appendix 3 - Section 9 - Other Safety Assessments

Appendix 3.9.1 – Other Safety Assessments: Vital Signs
- Treated Patients –

### Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Date | Height (cm) | Weight (kg) | Temperature (°C). | Route | Syst. B.P. (mmHg) | | Diast. B.P. (mmHg) | | Pulse<br>(bpm) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 35/M/W | Pretr. | ddmmmyyyy | XXX.X | XXX.X | XXX.X | XXXX | 170 | * | 100 | * | XXX |
| | | Cy 1 | ddmmmyyyy | | XXX.X | XXX.X | XXXX | 164 | * | XXX | | XXX |
| | | Cy 2 | ddmmmyyyy | | XXX.X | XXX.X | XXXX | XXX | | 110 | § | XXX |
| XXXX | | | | | | | | | | | | |

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.

(\*) Systolic Blood Pressure ≥140 mmHg or Diastolic Blood Pressure ≥ 90 mmHg.

(§) Increase from pretreatment: Systolic BP≥20; Diastolic BP≥10 mmHg.


[Program Path; Date/Time Produced; Date Data Extract]

<u>Programming notes</u>:

Sort by pt. no., study period, date.

## Appendix 3.9.2 – Other Safety Assessments: ECG - Treated Patients –

## Page by Regimen

| | Pt. No. | Age/Sex<br>/Race | Study Period | ECG Date | Ventricular<br>Rate<br>(bpm) | Tracing Abnormalities | Category | Specific Abnormality | Further Details |
|---|---|---|---|---|---|---|---|---|---|
| - | XXXX | 35/M/W | Pretr. | ddmmmyyyy | XXX | N | | | |
| | | | Cy 1 | ddmmmyyyy | xxx | Y | Rhythm<br>QRS | Sinus Tachicardia xxxxxxxxxxxx | |
| | | | Cy 2 | ddmmmyyyy | XXX | | | * XXXXXXX<br>XXXXXXX | |
| | | | Cy 3 | ddmmmyyyy<br>ddmmmyyyy | XXX | | | XXXXXXX<br>XXXXXXX | |
| | xxxx | xx/x/x | Pretr. | ddmmmyyyy | xxx | Y | ST-T<br>Wave | Other | xxxxxxx |
| | | | Cy 1 | ddmmmyyyy | | N | ••• | | |

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.

(\*) Specific Abnormality not present at pretreatment.


[Program Path; Date/Time Produced; Date Data Extract]

**Programming Notes:** 

Sort by pt. no., study period.

Appendix 3.9.3 – Other Safety Assessments: Visual Acuity and Funduscopic Examination - Treated Patients –

## Page by Regimen

| Study | | Cumulative | Date of | Snellen | Snellen | Date of | | |
|---|---|---|---|---|---|---|---|---|
| Pt. No. | Study<br>Period | Dose | Visual acuity | Equivalent | Equivalent | Funduscopic | Right Eye | Left Eye |
| 1 CHOU | | (mg) Assessment | | Right Eye | Left Eye | Examination | | |
| XXXX | Pretr. | | ddmmmyyyy | 20/xx | 20/xx | ddmmmyyyy | Normal | Normal |
| | Cy 1 | XXXX.X | ddmmmyyyy | 20/xx | 20/xx | ddmmmyyyy | Abnormal, clinically relevant | Abnormal, clinically relevant |
| | | | ddmmmyyyy | 20/xx | 20/xx | ddmmmyyyy | Abnormal, not clinically relevant | Abnormal, not clinically relevant |
| | Су ј | XXXX.X | ddmmmyyyy | | | ddmmmyyyy | Normal | Normal |
| | | XXXX.X | ddmmmyyyy | 20/xx | 20/xx | ddmmmyyyy | Abnormal, not clinically relevant | Abnormal, not clinically relevant |
| XXXX | | | | | | | | ••• |

Cumulative dose (mg): from treatment start up to end of relevant treatment cycle


[Program Path; Date/Time Produced; Date Data Extract]

Programming notes:

Sort by pt. no., study period.

#### Appendix 3.9.4 – Other Safety Assessments: Chest X-Ray - Treated Patients -

## Page by Regimen

| Pt. No | Age/Sex/Race | Date | Days<br>to/from<br>Tr. Start | Study<br>Period | Results |
|---|---|---|---|---|---|
| XXXX | 38/M/W | ddmmmyyyy | -1 | Pretr. | Normal |
| | | ddmmmyyyy | 4 | Cy 1 | Normal |
| | | ddmmmyyyy | 20 | | Abnormal; not clinically relevant |
| XXXX | xx/x/x | | | Pretr. | Abnormal; clinically relevant |
| | | • • • | | | ••• |

Only patients with chest x-ray performed are displayed

Race: W= White, B= Black, A= Asian, O= Not listed, N= Not allowed to ask per local regulation.

[Protocol No.; Study Description] [Program Path; Date/Time Produced; Date Data Extract]

Programming notes:

Sort by pt. no., date, study period.

## Appendix 3.9.5 – Other Safety Assessments: Pregnancy Test - Treated Patients –

## Page by Regimen

| Pt. No | Age/Sex/Race | Study<br>Period | Date | Method | Result | Reason for<br>Not Performing |
|---|---|---|---|---|---|---|
| XXXX | 38/F/W | Pretr. | | | | Surgically sterile |
| XXXX | 41/F/W | Pretr. | ddmmmyyyy | Serum | Negative | |
| XXXX | 43/F/W | ••• | ddmmmyyyy | Urine | Negative | |
| XXXX | 47/F/W | | ddmmmyyyy | Urine | Positive * | |
| XXXX | 57/F/W | | | | | Postmenopausal |

All female patients are displayed.

Race: W= White, B= Black, A= Asian, O= Not listed, N= Not allowed to ask per local regulation.

Result: Positive results are marked by a \*.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming notes:

Sort by pt. no., study period.

All female patients are to be displayed in the listing, including those for whom pregnancy test section is not present in the database.

#### Appendix 3.9.6 – Other Safety Assessments: Physical Examination - Treated Patients -

Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Physical Examination<br>(including neurological status<br>evaluation) Performed? | Date of Physical<br>Examination |
|---|---|---|---|---|
| XXXXXX | 35/M/W | Cy 1 | Y | ddmmmyyyy |
| | | Cy 2 | Y | ddmmmyyyy |
| | | Cy i | Y | ddmmmyyyy |
| XXXXXX | 50/M/W | Cy 1 | Y | ddmmmyyyy |
| | | Cv n | N | 2222 |

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.

[Protocol No.; Study Description] [Program Path; Date/Time Produced; Date Data Extract]

<u>Programming notes:</u>

Sort by pt. no., study period.

## Appendix 3 – Section 10 – Other Information

Appendix 3.10.1 - Other Information: Concomitant Medications - Treated Patients -

### Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Tr. Start<br>Date | Tr. Last<br>Date | Trade / Generic<br>Name | Reason for Use | Start Date | Stop Date | Ongoing at Final Visit (Y/N) | Duration (days) | Weeks<br>from<br>Tr. Start |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 35/M/W | ddmmmyyyy | ddmmmyyyy | xxxxxxxxxx | XXXXXXXXXXX | ddmmmyyyy | | Y | | XXX.X |
| | | | | XXXXXXXXXXX | XXXXXXXXXXX | ddmmmyyyy | ddmmmyyyy | | XXX | XXX.X |
| | | | | XXXXXXXXXXX | XXXXXXXXXXX | ddmmmyyyy | | Y | | XXX.X |
| XXXX | 50/M/W | ddmmmyyyy | ddmmmyyyy | XXXXXXXXXXX | XXXXXXXXXXX | ddmmmyyyy | ddmmmyyyy | | XXX | XXX.X |

Only patients with at least one concomitant medication are displayed

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.

Duration (days): from start date to stop date.

Weeks from Tr. Start: from treatment start date to start date of concomitant medication.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming notes:**

Sort by pt. no., start date.

Select only patients with concomitant medication='yes' or derived 'yes'
# Appendix 3.10.2 – Other Information: Concomitant Radiotherapies - Treated Patients –

## Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Tr. Start Date | Tr. Last<br>Date | Lesion Lesion<br>Number Description | % Bone<br>Marrow<br>Irradiated | Start Date | Stop Date | Duration (days) | Weeks<br>from<br>Tr. Start |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | 35/M/W | ddmmmyyyy | ddmmmyyyy | XXXX | XX.XX | ddmmmyyyy | | | XXX.X |
| | | | | XXXX | | ddmmmyyyy | ddmmmyyyy | XXX | XXX.X |
| | | | | | | ddmmmyyyy | | | XXX.X |
| XXXX | xx/x/x | ddmmmyyyy | ddmmmyyyy | | | ddmmmyyyy | ddmmmyyyy | XXX | XXX.X |

Only patients with at least one concomitant radiotherapy are displayed.

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation..

Duration (days): from start date to stop date.

Weeks from Tr. Start: from treatment start date to start date of concomitant radiotherapy.


[Program Path; Date/Time Produced; Date Data Extract]

# <u>Programming notes</u>:

Sort by pt no., start date.

Select only patients with concomitant radiotherapy = 'yes' or derived 'yes'.

# Appendix 3.10.3 – Other Information: Blood Derivatives - Treated Patients -

# Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Date | Weeks<br>from Tr.<br>Start | Type | Description | No. of Units |
|---|---|---|---|---|---|---|
| XXX | 35/M/W | ddmmmyyyy | XX.X | Whole Blood | | XX |
| | | | | Packed RBC | | |
| | | | | Packed WBC | | |
| XXX | xx/x/x | ddmmmyyyy | XX.X | Platelets | | |
| | | ddmmmyyyy | XX.X | Other | xxxxxxxxxxxxxxxxxx | ••• |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.. Weeks from Tr. Start: from treatment start date to date of blood derivatives.


[Program Path; Date/Time Produced; Date Data Extract]

<u>Programming Notes:</u>
Sort by pt. no, date.

Appendix 3.10.4 - Other Information: Other Anti-Tumor Therapies at Follow-up - Treated Patients –

#### Page by Regimen

| Pt.<br>No. | Age/Sex/Race | Visit | Start Date | Days from<br>Tr. Last Date | Description |
|---|---|---|---|---|---|
| XXXX | 35/M/W | FU-1 | ddmmmyyyy | XXX | xxxxxxxxxxxx |
| | | | ddmmmyyyy | XXX | XXXXXXXXXXXXXXX |
| | | | ddmmmyyyy | XXX | xxxxxxxxxxxxx |
| XXXX | xx/x/x | FU-2 | ddmmmyyyy | XXX | XXXXXXXXXXXXXX |

Only patients with at least one therapy are displayed.

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation..

Days from Tr. Last: from treatment last date to start date of anti-tumor therapy.


[Program Path; Date/Time Produced; Date Data Extract]

### **Programming Notes:**

Sort by pt. no., start date.

Select only patients with antitumor therapy ='yes' or derived 'yes'.

# Appendix 3.10.5 - Other Information: Physician's Comments - Treated Patients -

## Page by Regimen

| Pt. No. | Age/Sex/Race | Section | Visit | Page | Date | Comments |
|---|---|---|---|---|---|---|
| XXXX | 35/M/W | XXXXX | XXXXXXX | XX | ddmmmmyyyy | XXX XXXXX XXXXXXX XXXXXXXXXXXXXXXXXXXX |
| | | XXXXX | XXXXXXX | XX | ddmmmmyyyy | XXX XXXXX XXXXXXX XXXXXXXXXXXXXXXXXXXX |
| XXXX | xx/x/x | ••• | ••• | | ••• | |
| | | | ••• | | | ••• |
| XXXX | | | | | ••• | ••• |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation..


[Program Path; Date/Time Produced; Date Data Extract]

### **Programming Notes:**

Sort by pt. no., section, visit, page, date.

# **ADDITIONAL DISPLAYS**

Listing 3.3.1 – Patients Evaluability for Efficacy Analysis: Patients not Included in the Efficacy Analysis of Evaluable Patients - Enrolled Patients -

| Pt. No | First Dose<br>Date | Total Administered Dose in Cy1+Cy2 | Date of Last<br>Tumor<br>Assessment | Days<br>from<br>First<br>Dose | Date of<br>Death | Days<br>from<br>First<br>Dose | Reasons for Non-Evaluability |
|---|---|---|---|---|---|---|---|
| XXXX | | | ddmmmyyyy | | ddmmmyyyy | | Patient not treated |
| XXXX | ddmmmyyyy | XXX.X | ddmmmyyyy | -xx | | | Less than 80% of Intended Dose at Cy1+Cy2) / No tumor assessment at pretreatment |
| XXXX | ddmmmyyyy | xxx.x | | | | | No tumor assessment at pretreatment / No on treatment oncologic assessment nor death before (re)assessment |
| XXXX | ddmmmyyyy | XXX.X | ddmmmyyyy | XX | ddmmmyyyy | XX | No tumor assessment at pretreatment |


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Sort by patients no.. Report all reasons for non-evaluability.

Listing 3.4.1 – Demography and Pretreatment: Tumor History - Summary of Prior Antitumor Treatment Procedure - Treated Patients –

| Pt. No. | Age/Sex<br>/Race | Any Surgery? | Any Radiotherapy? | Any Systemic Therapy ? |
|---|---|---|---|---|
| XXXX | 38/M/W | Y | | Y |
| XXXX | xx/x/x | Y | | |
| XXXX | xx/x/x | | Y | |
| XXXX | xx/x/x | | | Y |
| XXXX | xx/x/x | Y | | |

Race: W= White, B= Black, A= Asian, O= Not Listed, N= Not Allowed to ask per local regulation.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming notes:

Sort by pt. no.

Listing 3.7.1 - Adverse Events: All Reported Adverse Events by AE MedDRA Preferred Term and Assessment Visit - Treated Patients -

| Pt.<br>No. | Adverse<br>Event | Study Period | Cycle<br>Start Date | CTC<br>Grade | Serious | Start Date | A.<br>P. | Stop Date | S.<br>P. | Rel.<br>to<br>Study<br>Proc. | Rel.<br>to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease | Action<br>Taken | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXXXXXXX | Pretr. | | 2 | | ddmmmyyyy | | ddmmmyyyy | | N | | N | | R |
| | | Cy 1 | ddmmmyyyy | 3 | | ddmmmyyyy | | | | | De | Y | D/C | NR |
| | | | | 4 | Y | | Y | | Y | | Pr | Y | D/C | R |
| | | Су х | ddmmmyyyy | | Y | | Y | ddmmmyyyy | | | | | PW | |
| | XXXXXXXXX | Cy 1 | ddmmmyyyy | 1 | | ddmmmyyyy | | ddmmmyyyy | | | | Y | No | NR |
| | | | | | | ddmmmyyyy | | | Y | | Po | ••• | | R |
| | | Cy x | ddmmmyyyy | | Y | | Y | ddmmmyyyy | | | | | | NR |
| XXXX | | ••• | | | | | | | | | | | | |

AP/SP: Already present/Still present.

Related to Study Treatment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.

Action Taken: No=None; D/C=Dose Delayed/Changed; PW=Drug Permanently Withdrawn.

Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by AE MedDRA Preferred Term, AE page no., AE seq no, pt. no., study period Include also records of End of Adverse Events Reporting Period and of Follow-up.

Listing 3.7.2 – Adverse Events: AEs with Possible/Probable/Definite Relationship to Study Treatment - Treated Patients -

| Pt. No | Study<br>Period | Cycle Start<br>Date | Adverse<br>Event | CTC<br>Grade | Serious | Start Date | A.<br>P. | Stop Date | S.<br>P. | Rel.<br>to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease | Action<br>Taken | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | Cy 1 | ddmmmyyyy | XXXXXXXXX | 1 | N | ddmmmyyyy | | ddmmmyyyy | | Po | N | | R |
| | | | XXXXXXXXX | 1 | N | | Y | | Y | Pr | N | | NR |
| | | | XXXXXXXXX | 2 | | | Y | ddmmmyyyy | | De | Y | | R |
| | Cy 2 | ddmmmyyyy | XXXXXXXXX | X | | | Y | | Y | Po | | No | NR |
| | | | XXXXXXXXX | | ••• | ddmmmyyyy | | | Y | De | N | No | NR |
| | | | xxxxxxxxx | 3 | Y | ddmmmyyyy | | ddmmmyyyy | | De | Y | D/C | R |

AP/SP: Already present/Still present.

Related to Study Treatment: Po=Possible, Pr=Probable, De=Definite.

Action Taken: No=None; D/C=Dose Delayed/Changed; PW=Drug Permanently Withdrawn.

Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Sort by pt. no., study period, AE MedDRA Preferred Term, AE page no., AE seq. no. Only AEs with possible/probable/definite relationship to study treatment are to be selected.

# Listing 3.7.3 – Adverse Events: AEs Leading to Dose Delay or Change - Treated Patients -

# Page by Regimen

| Pt. No | Study<br>Period | Cycle Start<br>Date | Adverse<br>Event | CTC<br>Grade | Serious | Start Date | A.<br>P. | Stop Date | S.<br>P. | Rel.<br>to<br>Study<br>Treat. | Rel. to<br>Study<br>Disease | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | Cy 1 | ddmmmyyyy | XXXXXXXXX | 1 | N | ddmmmyyyy | | ddmmmyyyy | | Po | N | R |
| | | | XXXXXXXXX | 1 | N | | Y | | Y | Pr | N | NR |
| | | | XXXXXXXXX | 2 | | | Y | ddmmmyyyy | | De | Y | R |
| | Cy 2 | ddmmmyyyy | XXXXXXXXX | X | | | Y | | Y | Po | | NR |
| | - | | XXXXXXXXX | | | ddmmmyyyy | | | Y | De | N | NR |
| | | | xxxxxxxxx | 3 | Y | ddmmmyyyy | | ddmmmyyyy | | De | Y | R |

Only AE occurrences at the time when Action Taken was Dose Delay or Change are displayed.

AP/SP: Already present/Still present.

Related to Study Treatment: No=Unrelated, Un=Unlikely, Po=Possible, Pr=Probable, De=Definite.

Outcome: R=Recovered; RS=Recovered with sequelae; D=Death; Un=Unknown; NR=Not recovered.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Sort by pt. no., study period, AE MedDRA Preferred Term, AE page no., AE seq. no..

Selct only the occurrences of AEs when variable Action Taken= 'Dose Delayed/Changed'.

Listing 3.8.1 - Laboratory Assessments: Hematology by Patient, Study Period and Laboratory Test
- Treated Patients –

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Cycle<br>Start Date | Date of Sampling | Study<br>Day | Lab. Test | Collected<br>Value | Collected<br>Unit | L/H | Converted<br>Value | Converted<br>Unit | CTC<br>Grade |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 52/F/W | Pretr. | ddmmmyyyy | ddmmmyyyy | -xx | Hemoglobin | XXX.XX | XXXX | L | XXX.XX | XXXX | X |
| | | | | | | Platelet | | | ••• | | | 3 * |
| | | | | | | WBC | ••• | ••• | • • • • | | ••• | 4 * |
| | | | | | | | | | ••• | | | |
| | | Cycle x | ddmmmyyyy | ddmmmyyyy | XX | Hemoglobin | | ••• | • • • | ••• | • • • | 2 |
| ••• | ••• | ••• | | | | Platelet | | | ••• | | | ••• |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

Converted Unit: either the unit reported in the NCI CTCAE v3.0 or the Conventional Unit, depending on the analyzed lab test.

CTC Grade - NCI CTCAE v3.0: N= Not Applicable, U= Unknown. The '\*' identifies the occurrence(s) of CTC grades= 3 or 4.

L/H: Below/Above Normal Limits.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by pt. no, study period, date of sampling, study day, lab test. If feasible lab test is to be ordered as per CRF appearance.

The listing must include all the hematological labs (including also the ones that are not listed in the NCI CTCAE v.3.0).

Each assessment (i.e. record) is to be displayed only if date is not missing or collected value is not missing.

Lisring 3.8.2 – Laboratory Assessments: Hematology by Laboratory Test, Patient and Study Periods with More than One Assessment - Treated Patients -

Page by Regimen /Laboratory Test: < Neutrophils >

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Cycle<br>Start Date | Cycle Total<br>Dose<br>(mg) | Date of Sampling | Study<br>Day | Collected<br>Value | Collected<br>Unit | L/H | Converted<br>Value | Converted<br>Unit | CTC<br>Grade |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 52/F/W | Pretr. | | | ddmmmyyyy | -XX | XXX.XX | XXXX | L | XXX.XX | XXXX | X |
| | | Су х | ddmmmyyyy | XXXX.XX | ddmmmyyyy | XX | ••• | ••• | | ••• | ••• | 3 * |
| | | | | | | XX | | ••• | • • • | ••• | ••• | 4 * |
| | | | | | | | | | • • • | | | |
| XXXX | | Pretr. | | | ddmmmyyyy | XX | | | • • • | | | 2 |
| | | | ••• | | | | | | | ••• | • • • | ••• |

Only study periods with more than one assessment for the test are displayed

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

Converted Unit: either the unit reported in the NCI CTCAE v3.0 or the Conventional Unit, depending on the analyzed lab test.

CTC Grade - NCI CTCAE v3.0: N= Not Applicable, U= Unknown. The '\*' identifies the occurrence(s) of CTC grades= 3 or 4.

L/H: Below/Above Normal Limits.


[Program Path; Date/Time Produced; Date Data Extract]

#### Programming Notes:

Sort by "page by variables", pt. no, study period, date of sampling, study day. If feasible lab test is to be ordered as per CRF appearance.

The listing must include all the hematological labs (including also the ones that are not listed in the NCI CTCAE v.3.0).

Each selected assessment (i.e. record) is to be displayed only if date is not missing or collected value is not missing.

Listing 3.8.3 – Laboratory Assessments: Hematology – Maximum CTC Grade by Laboratory Test, Patient and Time Window - Treated Patients –

Page by Regimen

#### Maximum CTC Grade at Laboratory Pt. All Cycle 1 Cycles >1 Pretr. Test No. Cycles Neutrophils 2 4 \* XXXX 2 \* 2 \* XXXX X XXXX X XXXX X X X X XXXX

Only lab. test included in the NCI CTCAE v3.0 document are displayed.

Pretreatment Value: the most recent value among the pretreatment assessment(s).

CTC Grade - NCI CTCAE v3.0: U= Unknown. The '\*' identifies CTC grades higher than Pretreatment grade.


[Program Path; Date/Time Produced; Date Data Extract]

#### <u>Programming Notes:</u>

Sort by lab test, pt. no. If feasible lab test is to be ordered as per CRF appearance.

Select collected lab tests listed in NCI CTCAE v3.0.

Listing 3.8.4 - Laboratory Assessments: Blood Chemistry by Patient, Study Period and Laboratory Test
- Treated Patients –

#### Page by Regimen

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Cycle<br>Start Date | Date of Sampling | Study<br>Day | Lab. Test | Collected<br>Value | Collected<br>Unit | d Collected<br>Lower Limi | Collected<br>Upper<br>Limit | L/H | Converted<br>Value | Converted<br>Unit | CTC<br>Grade |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 52/F/W | Pretr. | ddmmmyyyy | ddmmmyyyy | -xx | ALT | XXX.XX | XXXX | XXX.XX | XXX.XX | L | XXX.XX | XXXX | X |
| | | | | | | AST | ••• | | | | | | ••• | 3 * |
| | | | | | | Albumin | ••• | | | | | ••• | | 4 * |
| | | | | | | | | ••• | | | | | | ••• |
| | | Cycle x | ddmmmyyyy | ddmmmyyyy | XX | ALT | • • • | ••• | | | | | ••• | 2 |
| | | ••• | | | | AST | | • • • • | | | | | | |
| | | | ••• | ••• | | | | | | | | | ••• | |

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

Converted Unit: either the unit reported in the NCI CTCAE v3.0 or the Conventional Unit, depending on the analyzed lab test.

CTC Grade - NCI CTCAE v3.0: N= Not Applicable, U= Unknown. The '\*' identifies the occurrence(s) of CTC grades = 3 or 4.

L/H: Below/Above Normal Limits.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by pt. no, study period, date of sampling, study day, lab test. If feasible lab test is to be ordered as per CRF appearance.

The listing must include all the blood chemistry labs (including also the ones that are not listed in the NCI CTCAE v.3.0).

Each assessment (i.e. record) is to be displayed only if date is not missing or collected value is not missing.

Listing 3.8.5 – Laboratory Assessments: Blood Chemistry by Laboratory Test, Patient and Study Periods with More than One Assessment - Treated Patients -

Page by Regimen /Laboratory Test: < ALT >

| Pt.<br>No. | Age<br>/Sex<br>/Race | Study<br>Period | Cycle Start<br>Date | Cycle Total<br>Dose<br>(mg) | Date of Sampling | Study<br>Day | Collected<br>Value | Collected<br>Unit | Collected<br>Lower<br>Limit | Collected<br>Upper<br>Limit | L/H | Converted<br>Value | Converted<br>Unit | CTC<br>Grade |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | 52/F/W | Pretr. | | | ddmmmyyyy | - XX | XXX.XX | XXX.XX | XXX.XX | XXX | L | XXX.XX | XXXX | N |
| | | | | | | | XXX.XX | XXX.XX | XXX.XX | XXX | | | | N |
| | | Cy x | ddmmmyyyy | XXXX.XX | ddmmmyyyy | XX | XXX.XX | XXX.XX | XXX.XX | XXX | Н | ••• | | 3* |
| | | | | | | | | | | ••• | | | | |
| | | | | | | | | | | | • • • • | ••• | | |
| | | | | | ddmmmyyyy | XX | | | | | L | | | 4* |
| ••• | | ••• | ••• | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | | | |

Only study periods with more than one assessment for the test are displayed

Race: W=White, B=Black, A=Asian, O=Not listed, N=Not allowed to ask per local regulation.

Converted Unit: either the unit reported in the NCI CTCAE v3.0 or the Conventional Unit, depending on the analyzed lab test.

CTC Grade - NCI CTCAE v3.0: N= Not Applicable, U= Unknown. The '\*' identifies the occurrence(s) of CTC grades= 3 or 4.

L/H: Below/Above Normal Limits.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by "page by variables", pt. no, study period, date of sampling, study day.

If feasible lab test is to be ordered as per CRF appearance.

The listing must include all the biochemistry labs (including also the ones that are not listed in the NCI CTCAE v.3.0).

Each selected assessment (i.e. record) is to be displayed only if date is not missing or collected value is not missing.

Listing 3.8.6 – Laboratory Assessments: Blood Chemistry - Maximum CTC Grade by Laboratory Test, Patient and Time Window (Part I)

- Treated Patients -

Page by Regimen

| | | | at | | |
|---|---|---|---|---|---|
| Laboratory<br>Test | Pt.<br>No. | Pretr. | Cycle 1 | Cycles >1 | All<br>Cycles |
| ALT | XXXX | 3 | 2 | 4 * | 4 * |
| | XXXX | 1 | 2 * | 1 | 2 * |
| | XXXX | X | X | X | X |
| | XXXX | X | X | X | X |
| | XXXX | X | X | X | X |
| Albumin | XXXX | 0 | 1* | 2* | 2* |

Only lab. tests included in the NCI CTCAE v3.0 document and whose abnormality is determined by one-way modifications only, are displayed. Pretreatment Value: the most recent value among the pretreatment assessment(s).

CTC Grade - NCI CTCAE v3.0: U= Unknown. The '\*' identifies CTC grades higher than Pretreatment grade.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by lab test, pt. no. If feasible lab test is to be ordered as per CRF appearance.

Select collected lab tests listed in NCI CTCAE v3.0.

Listing 3.8.7 – Laboratory Assessments: Blood Chemistry - Maximum CTC Grade by Laboratory Test, Patient and Time Window (Part II)

- Treated Patients -

#### Page by Regimen

| | _ | Maximum CTC Grade at | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory<br>Test | Pt.<br>No. | Pretreatment | | Cycle 1 | | Cycles >1 | | | All Cycles | | | | |
| | - | L | N | Н | L | N | Н | L | N | Н | L | N | Н |
| Calcium | XXXX | | 0 | | 2 | | | 2 | | 1 | 2 | | 1 |
| | XXXX | | 0 | | | 0 | | | | 3 | | | 3 |
| | XXXX | | 0 | | | 0 | | | 0 | | | 0 | |
| | XXXX | 1 | | | 2 | | | 3 | | | 3 | | |
| | XXXX | | | | | | | | | | | | |
| Sodium | XXXX | | | | | | | | | | | | |

Only lab. tests included in the NCI CTCAE v3.0 document and whose abnormality is determined by two-way modifications (L = value lower than normal range, H = value higher than normal range, N= value within normal range), are displayed.

Pretreatment Value: the most recent value among the pretreatment assessment(s).

CTC Grade - NCI CTCAE v3.0: U= Unknown.


[Program Path; Date/Time Produced; Date Data Extract]

#### **Programming Notes:**

Sort by lab test, pt. no. If feasible lab test is to be ordered as per CRF appearance.

Select collected lab tests listed in NCI CTCAE v3.0 for which both 'hyper' and 'hypo' grading is provided. For this study: Magnesium, Potassium, Sodium.

# **REVISION HISTORY**

| Version | Date | Reviewed by: (Printed name) | Reason for change |
|---|---|---|---|
| 1.0 | 22 April 2013 | n.a. | First release of the document |

Reviewed and Approved by:

| Role | Printed Name | Signature | Date |
|--------------|---------------------|-----------|------|
| Statistician | Anna Petroccione | | |
| CL | Marcella Martignoni | | |